CLINICAL TRIAL: NCT06995586
Title: The Synergistic Action of Vitamins and Dietary Supplements in Patients With Coronary Artery Bypass Grafting for Improving the Quality of Healthcare Delivery.
Brief Title: Dietary Supplements in Patients With Coronary Artery Bypass Grafting for Improving the Quality of Healthcare Delivery.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicosia General Hospital (Other)
Collaborators: University of Cyprus (Other); AVVA Pharmaceuticals Ltd. (Industry)
Responsible Party: Principal Investigator, Athanasios Athanasiou, Cardiothoracic Surgeon (CTS), MD, MSc, MSc, MPA, PhD(cand.), Nicosia General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 36/22; Research Proposal: RP/2022/35 (Other: Cyprus National Bioethics Committe (EU))
Record Dates: First submitted 2025-04-25; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cardio-pulmonary Bypass; Cardiovascular Diseases; Omega-3 Polyunsaturated Fatty Acids; Omega-3 Supplementation; Vitamin C; Supplements; Postoperative Depression; Antioxidants; Lactulose; Postoperative; Optimal Medical Therapy; CABG; Coronary Artery Bypass Grafting; Prebiotics
Keywords: Cardio-pulmonary Bypass; Cardiovascular Diseases; Omega-3 polyunsaturated fatty acids; Vitamin C; Antioxidants; Lactulose; Omega-3 supplementation; Supplements; postoperative; Optimal Medical Therapy; CABG; Coronary Artery Bypass Grafting; postoperative depression; Lignin; adsorbent; prebiotics
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ascorbic Acid; Lignin; Lactulose

STUDY DESIGN:
Intervention Model Description: This is a randomized and controlled trial with an intervention group that will be administered orally daily in addition to the Optimal Medical Therapy (OMT), namely 1000 mg Vitamin C, 840 mg EPO/DHA, 2130 mg Lignin & 720 mg Lactulose and a control group that will receive only the OMT.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (OMT & Supplements) (Experimental): This is a randomized and controlled trial with an intervention group that will be administered orally daily 1000 mg Vitamin C, 840 mg EPO/DHA, 2130 mg Lignin & 720 mg Lactulose in addition to the Optimal Medical Therapy (OMT).
  Interventions: Dietary Supplement: Vitamin C, Omega 3 PUFA (EPO/DHA), Lignin, Lactulose
- Control group (OMT) (No Intervention): This is a randomized and controlled trial with an intervention group and a control group that will receive only the Optimal Medical Therapy (OMT).

INTERVENTIONS:
Dietary Supplement: Vitamin C, Omega 3 PUFA (EPO/DHA), Lignin, Lactulose — This is a randomized and controlled trial with an intervention group that will be administered orally daily in addition to the Optimal Medical Therapy (OMT), namely 1000 mg Vitamin C, 840 mg EPO/DHA, 2130 mg Lignin & 720 mg Lactulose and a control group that will receive only the OMT.
  Arms: Intervention group (OMT & Supplements)

SUMMARY:
Cardiovascular disease (CVD) remains the leading cause of death worldwide. Prevention of CAD by targeting modifiable factors remains a key public health priority. L-Ascorbic Acid (Vitamin C - Vit. C) and Omega 3 fatty acids, Eicosapentaenoic / Docosahexaenoic Acid (EPO/DHA), powerful but also necessary antioxidants for the human body, after observational studies as well as randomized studies seem to have a beneficial effect in the direction of the prevention of CVD with pleiotropic mechanisms. Lignin, a polymer of plant origin that is considered a dietary fiber, has a developed porous structure and can retain exogenous and endogenous toxins, and pathogenic microorganisms. Lactulose considered a prebiotic provides a selective substrate for the metabolism of saccharolytic bacteria with bifidogenic activity and multiple benefits to the host's gut health. Coronary artery bypass grafting (CABG) is an established surgical intervention and treatment of symptoms of myocardial ischemia that improves patient survival Optimal Medical Therapy (OMT) after coronary arterial bypass grafting (CABG) as described in current clinical practice could be made even better by the addition of these beneficial food supplements.

A randomized controlled trial is proposed in an intervention group of 54 post-CABG patients who will be given daily orally in addition to the usual medication, 1000 mg Vitamin C, 840 mg EPO/DHA, 2130 mg Lignin & 720 mg Lactulose and a control group of 54 patients (Control Group) in which only usual medication will be administered. The intervention will take place from the 15th postoperative day when CAGB patients are discharged and lasts for 2.5 months (10 weeks) postoperatively. The data will be collected on the 15th, 80-90th postop day in 6 months and 12 months postop and then the statistical analysis of the data will be performed. Considering the number of CABG surgeries performed electively in our clinic, this study is expected to be completed in approximately 2-3 years from the day of initiation.

The expected knowledge through the expected results such as these will emerge from this study is the potentially beneficial effect of our food supplements administration (intervention), i.e. Vitamin C, EPO/DHA, Lignin & Lactulose, on the postoperative course of our patients. Some degree of improvement in the well-being and clinical picture of our patients postoperatively is expected, which will be thoroughly investigated in each phase of the study.

DETAILED DESCRIPTION:
Background: Cardiovascular disease (CVD) remains the leading cause of death worldwide. CVD is the result of disorders of the heart and blood vessels and includes cerebrovascular disease, coronary artery disease (CAD) and peripheral arterial disease. The main mechanism believed to cause CAD is atherosclerosis, in which the arteries become narrowed by plaques or atheroma. While arteries can naturally become harder and narrower with age, this process can be accelerated by factors such as smoking, high cholesterol, high blood pressure, obesity, a sedentary lifestyle and ethnicity. Prevention of CAD by targeting modifiable factors remains a key public health priority. Diet plays an important role in the etiology of many chronic diseases including CAD, thus contributing to a significant geographic variability in morbidity and mortality rates between different countries and populations worldwide. A number of dietary factors have been found to be associated with CAD risk and can be modified to reduce CAD risk with interventions aimed at CAD prevention and management. L-Ascorbic Acid (Vitamin C - Vit. C) and Omega 3 fatty acids, Eicosapentaenoic / Docosahexaenoic Acid (EPO/DHA), powerful but also necessary antioxidants for the human body, after observational studies as well as randomized studies seem to have a beneficial effect in the direction of the prevention of CVD with pleiotropic mechanisms. Lignin, a polymer of plant origin that is considered a dietary fiber, has a developed porous structure and can retain exogenous and endogenous toxins, and pathogenic microorganisms. Lactulose considered a prebiotic provides a selective substrate for the metabolism of saccharolytic bacteria with bifidogenic activity and multiple benefits to the host's gut health.

Objectives of the study: Our work, which is unique in its kind, is expected to highlight and help establish the administration of the proposed formulations (Vitamin C, EPO/DHA, Lignin, Lactulose) as an integral part of optimal medical therapy (OMT) after interventions in the coronary vessels. It will also form the basis for further research regarding the combined physiological mechanisms of action of the vitamins in question (Vitamin C, EPO/DHA, Lignin, Lactulose) both at the histological and cellular level.

Description of methods including collection and analysis: This is a randomized and controlled trial with an intervention group that will be administered orally daily in addition to the OMT, namely 1000 mg Vitamin C, 840 mg EPO/DHA, 2130 mg Lignin & 720 mg Lactulose and a control group that will receive only the OMT. The intervention will take place from the 15th postoperative day (POD) when CAGB patients are discharged and lasts for 2.5 months (10 weeks) PO. The data will be collected on the 15th, 80-90th POD in 6 months and 12 months PO and then the statistical analysis of the data will be performed. Considering the number of CABG surgeries performed electively in our clinic, this study is expected to be completed in approximately 3 years from the day of its initiation. The subjects will be people 40-80 years old, with coronary artery disease, and mental clarity without any psychiatric, neurological or motor disorder who will undergo Coronary Aortic Bypass (CABG) in our clinic (Public Cardiothoracic Surgery clinic in Nicosia General Hospital) and will be randomized into 2 groups (intervention group and control group). A total of at least 108 subjects are required for both groups (54 in each group). In this way, a 40% incidence could be detected in the control group with a 16% incidence in the intervention group (Vitamin C, EPO/DHA, Lignin, Lactulose), i.e. a reduction of around 60% (Alpha 5%, Beta 20%, Power 80%). Once informed consent and written consent have been obtained from a subject and satisfactory inclusion and exclusion criteria have been verified, the individual will be assigned to a group and undergo physical examinations and laboratory blood tests to confirm their status. Each subject will be randomly assigned to each group using a random number generator that assigns each subject to each group in a blinded fashion. A questionnaire asking patients about their experience and opinion of the quality of our services and the patients' quality of life before and after surgery will also be distributed, as well as a consent form to enroll in the study. The data will be collected during the 1st to 4th PO appointment namely the 15th POD, the 80-90th POD in 6 months and 12 months PO in a database on a computer of our hospital and then the statistical analysis of the data will be carried out with the appropriate software. All appropriate parametric and non-parametric statistical analyzes will be performed accordingly (X2 test, Logistic Regression, Linear Regression, Analysis of Variance (ANOVA), Log Rank test, Cox hazard model, ROC curve, etc.). Appropriate statistical analysis software (IBM® SPSS®) will be applied and in addition, assistance from a specialist statistician will be requested for highly specialized analyses.

Project Innovation and Originality: OMT postoperatively (PO) is subject to improvement. One of these promising improvements is the addition of (Vitamin C, EPO/DHA, Lignin, Lactulose) proposed by the present study, for which the research in question is being carried out. As far as we know, the proposed study is the first of its kind internationally that studies the combined action of these 4 factors together, which makes it unique. Some degree of improvement in the well-being and clinical picture of our patients PO is expected, which will be thoroughly investigated in each phase of the study. In this way, both the theoretical framework around PO treatment and the clinical practice itself in which we propose to introduce the aforesaid complementary treatment will be improved.

Dissemination of findings: The results of our study, which is part of Dr. Athanasiou's doctoral thesis at the Open University of Cyprus under the supervision of Dr. Soteriades, will be shared and published both in the domestic and international scientific press and will be freely accessible through the servers of the Open University of Cyprus. There will be no royalties and no charge for acquiring the original work and publications.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be people 40-80 years old, with coronary artery disease, and mental clarity who will undergo Coronary Aortic Bypass (CABG) in our clinic (Public Cardiothoracic Surgery clinic in Nicosia General Hospital) and will be randomized into 2 groups (intervention group and control group).
* Signed consent form
* Ability to adhere to the protocol

Exclusion Criteria:

* Any psychiatric, neurological or motor disorder.
* Hypersensitivity to the components of the supplement.
* Combined Cardiac Surgery other than CABG and valve or aortic
* Concurrent participation in other clinical trials.
* Previous use of any probiotics, prebiotics, adsorbent dietary supplements, Vitamin C and/or Omega 3 fatty acids.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative decrease in morbidity/mortality associated with our intervention complementary to OMT (Vit C, n-3 PUFA, Lignin and Lactulose) | The data will be collected on the 15th, 80-90th postop day (POD) in 6 months and 12 months PO and then the statistical analysis of the data will be performed. This study is expected to be completed in approximately 3 years from the day of its initiation.
  Optimal Medical Therapy (OMT) postoperatively (PO) is subject to improvement. One of these promising improvements is the addition of (Vitamin C, EPO/DHA, Lignin, Lactulose) proposed by the present study, for which the research in question is being carried out. As far as we know, the proposed study is the first of its kind internationally that studies the combined action of these 4 factors together, which makes it unique. Some degree of improvement in the well-being and clinical picture of our patients PO is expected, which will be thoroughly investigated in each phase of the study. In this way, both the theoretical framework around PO treatment and the clinical practice itself in which we propose to introduce the aforesaid complementary treatment will be improved.

SECONDARY OUTCOMES:
Overall Quality Assesment. Assesment of the quality of the service provided to the patients & overall quality of life of our patients postoperatively. | The data will be collected on the 15th, 80-90th postop day (POD) in 6 months and 12 months PO and then the statistical analysis of the data will be performed. This study is expected to be completed in approximately 3 years from the day of its initiation.
  There will be questionnaires assessing the perceived quality of our health service to the patient as well as objective/actual measurements about the overall quality of life of our patients postoperatively. These data will be assessed in 4 time points postoperatively.
Postoperative Mental Status of the patients. | The data will be collected on the 15th, 80-90th postop day (POD) in 6 months and 12 months PO and then the statistical analysis of the data will be performed. This study is expected to be completed in approximately 3 years from the day of its initiation.
  There will be an internationally standardized questionnaire, namely "The Center for Epidemiologic Studies-Depression scale (CES-D Scale), about the mental status of our patients and it will be assessed in 4 time points postoperatively. The CES-D measures a well-being/depression continuum in adolescents, adults, and older adults. The CES-D total score provides an indication of depressive symptom severity that is based on a combination of the presence/absence of depressive experiences and the presence/absence of well-being. Possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology.

OTHER OUTCOMES:
Full blood count (FBC) examination postoperatively during the follow up period. | The data will be collected on the 15th, 80-90th postop day (POD) in 6 months and 12 months PO and then the statistical analysis of the data will be performed. This study is expected to be completed in approximately 3 years from the day of its initiation.
  Individuals who participate in this study will receive additional follow-up postoperatively for one year according to the protocol and have full blood count (FBC) blood test.
Biochemical analysis postoperatively during the follow up period. | The data will be collected on the 15th, 80-90th postop day (POD) in 6 months and 12 months PO and then the statistical analysis of the data will be performed. This study is expected to be completed in approximately 3 years from the day of its initiation.
  Individuals who participate in this study will receive additional follow-up postoperatively for one year according to the protocol and have biochemical analysis blood test.
C reactive protein (CRP) examination postoperatively during the follow up period. | The data will be collected on the 15th, 80-90th postop day (POD) in 6 months and 12 months PO and then the statistical analysis of the data will be performed. This study is expected to be completed in approximately 3 years from the day of its initiation.
  Individuals who participate in this study will receive additional follow-up postoperatively for one year according to the protocol and have C reactive protein (CRP) examination blood test.
Echocardiographic examination postoperatively during the follow up period. | The data will be collected on the 80-90th postop day (POD) in 6 months and 12 months PO and then the statistical analysis of the data will be performed. This study is expected to be completed in approximately 3 years from the day of its initiation.
  Individuals who participate in this study will receive additional follow-up postoperatively for one year according to the protocol and have heart Echocardiography.
Radiologic examinations postoperatively during the follow up period. | The data will be collected on the 15th, 80-90th postop day (POD) in 6 months and 12 months PO and then the statistical analysis of the data will be performed. This study is expected to be completed in approximately 3 years from the day of its initiation.
  Individuals who participate in this study will receive additional follow-up postoperatively for one year according to the protocol and have radiological examinations with a Chest X-ray.
Physical examination (weight measurement) postoperatively during the follow up period. | The data will be collected on the 15th, 80-90th postop day (POD) in 6 months and 12 months PO and then the statistical analysis of the data will be performed. This study is expected to be completed in approximately 3 years from the day of its initiation.
  Individuals who participate in this study will receive additional follow-up postoperatively for one year according to the protocol and have on site weight measurement in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Elpidoforos S. Soteriades, MD, Ass Prof, Study Chair — Open University of Cyprus; Athanasios D. Athanasiou, MD, MSc, MPA, Principal Investigator — Nicosia General Hospital; Elpidoforos S. Soteriades, MD, Ass Prof, Study Director — Open University of Cyprus
Locations (1):
- Nicosia General Hospital, Stróvolos, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miloyan, B., Eaton, W.W. (2021). The Center for Epidemiologic Studies Depression (CES-D) Scale. In: Gu, D., Dupre, M.E. (eds) Encyclopedia of Gerontology and Population Aging. Springer, Cham. https://doi.org/10.1007/978-3-030-22009-9_416
- [Background] Siddaway AP, Wood AM, Taylor PJ. The Center for Epidemiologic Studies-Depression (CES-D) scale measures a continuum from well-being to depression: Testing two key predictions of positive clinical psychology. J Affect Disord. 2017 Apr 15;213:180-186. doi: 10.1016/j.jad.2017.02.015. Epub 2017 Feb 20. PMID 28254608
- [Background] Zhao YC, Wang CC, Yang JY, Li XY, Yanagita T, Xue CH, Zhang TT, Wang YM. N-3 PUFA Deficiency from Early Life to Adulthood Exacerbated Susceptibility to Reactive Oxygen Species-Induced Testicular Dysfunction in Adult Mice. J Agric Food Chem. 2023 May 10;71(18):6908-6919. doi: 10.1021/acs.jafc.2c07328. Epub 2023 Apr 25. PMID 37098125
- [Background] Madore C, Nadjar A, Delpech JC, Sere A, Aubert A, Portal C, Joffre C, Laye S. Nutritional n-3 PUFAs deficiency during perinatal periods alters brain innate immune system and neuronal plasticity-associated genes. Brain Behav Immun. 2014 Oct;41:22-31. doi: 10.1016/j.bbi.2014.03.021. Epub 2014 Apr 13. PMID 24735929
- [Background] Cole GM, Ma QL, Frautschy SA. Omega-3 fatty acids and dementia. Prostaglandins Leukot Essent Fatty Acids. 2009 Aug-Sep;81(2-3):213-21. doi: 10.1016/j.plefa.2009.05.015. Epub 2009 Jun 12. PMID 19523795
- [Background] Delpech JC, Thomazeau A, Madore C, Bosch-Bouju C, Larrieu T, Lacabanne C, Remus-Borel J, Aubert A, Joffre C, Nadjar A, Laye S. Dietary n-3 PUFAs Deficiency Increases Vulnerability to Inflammation-Induced Spatial Memory Impairment. Neuropsychopharmacology. 2015 Nov;40(12):2774-87. doi: 10.1038/npp.2015.127. Epub 2015 May 7. PMID 25948102
- [Background] Aid S, Vancassel S, Poumes-Ballihaut C, Chalon S, Guesnet P, Lavialle M. Effect of a diet-induced n-3 PUFA depletion on cholinergic parameters in the rat hippocampus. J Lipid Res. 2003 Aug;44(8):1545-51. doi: 10.1194/jlr.M300079-JLR200. Epub 2003 May 16. PMID 12754277
- [Background] Belkouch M, Hachem M, Elgot A, Lo Van A, Picq M, Guichardant M, Lagarde M, Bernoud-Hubac N. The pleiotropic effects of omega-3 docosahexaenoic acid on the hallmarks of Alzheimer's disease. J Nutr Biochem. 2016 Dec;38:1-11. doi: 10.1016/j.jnutbio.2016.03.002. Epub 2016 Mar 24. PMID 27825512
- [Background] McNamara RK, Almeida DM. Omega-3 Polyunsaturated Fatty Acid Deficiency and Progressive Neuropathology in Psychiatric Disorders: A Review of Translational Evidence and Candidate Mechanisms. Harv Rev Psychiatry. 2019 Mar/Apr;27(2):94-107. doi: 10.1097/HRP.0000000000000199. PMID 30633010
- [Background] Palacios-Pelaez R, Lukiw WJ, Bazan NG. Omega-3 essential fatty acids modulate initiation and progression of neurodegenerative disease. Mol Neurobiol. 2010 Jun;41(2-3):367-74. doi: 10.1007/s12035-010-8139-z. Epub 2010 May 14. PMID 20467837
- [Background] Leyrolle Q, Decoeur F, Dejean C, Briere G, Leon S, Bakoyiannis I, Baroux E, Sterley TL, Bosch-Bouju C, Morel L, Amadieu C, Lecours C, St-Pierre MK, Bordeleau M, De Smedt-Peyrusse V, Sere A, Schwendimann L, Gregoire S, Bretillon L, Acar N, Joffre C, Ferreira G, Uricaru R, Thebault P, Gressens P, Tremblay ME, Laye S, Nadjar A. N-3 PUFA deficiency disrupts oligodendrocyte maturation and myelin integrity during brain development. Glia. 2022 Jan;70(1):50-70. doi: 10.1002/glia.24088. Epub 2021 Sep 14. PMID 34519378
- [Background] Wang DD, Wu F, Zhang LY, Zhao YC, Wang CC, Xue CH, Yanagita T, Zhang TT, Wang YM. Effects of dietary n-3 PUFA levels in early life on susceptibility to high-fat-diet-induced metabolic syndrome in adult mice. J Nutr Biochem. 2021 Mar;89:108578. doi: 10.1016/j.jnutbio.2020.108578. Epub 2020 Dec 31. PMID 33388352
- [Background] Zou HY, Zhang HJ, Zhao YC, Li XY, Wang YM, Zhang TT, Xue CH. N-3 PUFA Deficiency Aggravates Streptozotocin-Induced Pancreatic Injury in Mice but Dietary Supplementation with DHA/EPA Protects the Pancreas via Suppressing Inflammation, Oxidative Stress and Apoptosis. Mar Drugs. 2023 Jan 1;21(1):39. doi: 10.3390/md21010039. PMID 36662212
- [Background] Ramirez JL, Zahner GJ, Spaulding KA, et al. HHS Public Access. 2020;54:211-19.
- [Background] Catry E, Neyrinck AM, Lobysheva I, Pachikian BD, Van Hul M, Cani PD, Dessy C, Delzenne NM. Nutritional depletion in n-3 PUFA in apoE knock-out mice: A new model of endothelial dysfunction associated with fatty liver disease. Mol Nutr Food Res. 2016 Oct;60(10):2198-2207. doi: 10.1002/mnfr.201500930. Epub 2016 Jun 1. PMID 27136390
- [Background] Danaei G, Ding EL, Mozaffarian D, Taylor B, Rehm J, Murray CJ, Ezzati M. The preventable causes of death in the United States: comparative risk assessment of dietary, lifestyle, and metabolic risk factors. PLoS Med. 2009 Apr 28;6(4):e1000058. doi: 10.1371/journal.pmed.1000058. Epub 2009 Apr 28. PMID 19399161
- [Background] Robertson RC, Seira Oriach C, Murphy K, Moloney GM, Cryan JF, Dinan TG, Ross RP, Stanton C. Deficiency of essential dietary n-3 PUFA disrupts the caecal microbiome and metabolome in mice. Br J Nutr. 2017 Dec;118(11):959-970. doi: 10.1017/S0007114517002999. Epub 2017 Nov 27. PMID 29173237
- [Background] Hutchins-Wiese HL, Picho K, Watkins BA, Li Y, Tannenbaum S, Claffey K, Kenny AM. High-dose eicosapentaenoic acid and docosahexaenoic acid supplementation reduces bone resorption in postmenopausal breast cancer survivors on aromatase inhibitors: a pilot study. Nutr Cancer. 2014;66(1):68-76. doi: 10.1080/01635581.2014.847964. Epub 2013 Nov 25. PMID 24274259
- [Background] Mocellin MC, de Quadros Camargo C, de Souza Fabre ME, et al. Fish oil effects on quality of life, body weight and free fat mass change in gastrointestinal cancer patients undergoing chemotherapy: a triple blind, randomized clinical trial. J Funct Foods 2017;31:113-22.
- [Background] Takezaki T, Inoue M, Kataoka H, Ikeda S, Yoshida M, Ohashi Y, Tajima K, Tominaga S. Diet and lung cancer risk from a 14-year population-based prospective study in Japan: with special reference to fish consumption. Nutr Cancer. 2003;45(2):160-7. doi: 10.1207/S15327914NC4502_04. PMID 12881009
- [Background] Patterson RE, Flatt SW, Newman VA, Natarajan L, Rock CL, Thomson CA, Caan BJ, Parker BA, Pierce JP. Marine fatty acid intake is associated with breast cancer prognosis. J Nutr. 2011 Feb;141(2):201-6. doi: 10.3945/jn.110.128777. Epub 2010 Dec 22. PMID 21178081
- [Background] Pan M, Zhao F, Xie B, Wu H, Zhang S, Ye C, Guan Z, Kang L, Zhang Y, Zhou X, Lei Y, Wang Q, Wang L, Yang F, Zhao C, Qu J, Zhou X. Dietary omega-3 polyunsaturated fatty acids are protective for myopia. Proc Natl Acad Sci U S A. 2021 Oct 26;118(43):e2104689118. doi: 10.1073/pnas.2104689118. PMID 34675076
- [Background] Sala-Vila A, Diaz-Lopez A, Valls-Pedret C, Cofan M, Garcia-Layana A, Lamuela-Raventos RM, Castaner O, Zanon-Moreno V, Martinez-Gonzalez MA, Toledo E, Basora J, Salas-Salvado J, Corella D, Gomez-Gracia E, Fiol M, Estruch R, Lapetra J, Fito M, Aros F, Serra-Majem L, Pinto X, Ros E; Prevencion con Dieta Mediterranea (PREDIMED) Investigators. Dietary Marine omega-3 Fatty Acids and Incident Sight-Threatening Retinopathy in Middle-Aged and Older Individuals With Type 2 Diabetes: Prospective Investigation From the PREDIMED Trial. JAMA Ophthalmol. 2016 Oct 1;134(10):1142-1149. doi: 10.1001/jamaophthalmol.2016.2906. PMID 27541690
- [Background] Balic A, Vlasic D, Zuzul K, Marinovic B, Bukvic Mokos Z. Omega-3 Versus Omega-6 Polyunsaturated Fatty Acids in the Prevention and Treatment of Inflammatory Skin Diseases. Int J Mol Sci. 2020 Jan 23;21(3):741. doi: 10.3390/ijms21030741. PMID 31979308
- [Background] Kim HH, Cho S, Lee S, Kim KH, Cho KH, Eun HC, Chung JH. Photoprotective and anti-skin-aging effects of eicosapentaenoic acid in human skin in vivo. J Lipid Res. 2006 May;47(5):921-30. doi: 10.1194/jlr.M500420-JLR200. Epub 2006 Feb 7. PMID 16467281
- [Background] Giudetti AM, Cagnazzo R. Beneficial effects of n-3 PUFA on chronic airway inflammatory diseases. Prostaglandins Other Lipid Mediat. 2012 Dec;99(3-4):57-67. doi: 10.1016/j.prostaglandins.2012.09.006. Epub 2012 Oct 11. PMID 23064030
- [Background] Pastor N, Soler B, Mitmesser SH, Ferguson P, Lifschitz C. Infants fed docosahexaenoic acid- and arachidonic acid-supplemented formula have decreased incidence of bronchiolitis/bronchitis the first year of life. Clin Pediatr (Phila). 2006 Nov;45(9):850-5. doi: 10.1177/1073858406289801. PMID 17041174
- [Background] Duttaroy AK, Basak S. Maternal dietary fatty acids and their roles in human placental development. Prostaglandins Leukot Essent Fatty Acids. 2020 Apr;155:102080. doi: 10.1016/j.plefa.2020.102080. Epub 2020 Feb 21. PMID 32120190
- [Background] Lucas M, Asselin G, Merette C, Poulin MJ, Dodin S. Effects of ethyl-eicosapentaenoic acid omega-3 fatty acid supplementation on hot flashes and quality of life among middle-aged women: a double-blind, placebo-controlled, randomized clinical trial. Menopause. 2009 Mar-Apr;16(2):357-66. doi: 10.1097/gme.0b013e3181865386. PMID 19034052
- [Background] Shek LP, Chong MF, Lim JY, Soh SE, Chong YS. Role of dietary long-chain polyunsaturated fatty acids in infant allergies and respiratory diseases. Clin Dev Immunol. 2012;2012:730568. doi: 10.1155/2012/730568. Epub 2012 Aug 28. PMID 23049602
- [Background] Stanhiser J, Jukic AMZ, McConnaughey DR, Steiner AZ. Omega-3 fatty acid supplementation and fecundability. Hum Reprod. 2022 May 3;37(5):1037-1046. doi: 10.1093/humrep/deac027. PMID 35147198
- [Background] Behboudi-Gandevani S, Hariri FZ, Moghaddam-Banaem L. The effect of omega 3 fatty acid supplementation on premenstrual syndrome and health-related quality of life: a randomized clinical trial. J Psychosom Obstet Gynaecol. 2018 Dec;39(4):266-272. doi: 10.1080/0167482X.2017.1348496. Epub 2017 Jul 14. PMID 28707491
- [Background] Donadio JV, Grande JP. The role of fish oil/omega-3 fatty acids in the treatment of IgA nephropathy. Semin Nephrol. 2004 May;24(3):225-43. doi: 10.1016/j.semnephrol.2004.01.004. PMID 15156528
- [Background] Kiecolt-Glaser JK, Belury MA, Andridge R, Malarkey WB, Glaser R. Omega-3 supplementation lowers inflammation and anxiety in medical students: a randomized controlled trial. Brain Behav Immun. 2011 Nov;25(8):1725-34. doi: 10.1016/j.bbi.2011.07.229. Epub 2011 Jul 19. PMID 21784145
- [Background] Doaei S, Bourbour F, Teymoori Z, Jafari F, Kalantari N, Abbas Torki S, Ashoori N, Nemat Gorgani S, Gholamalizadeh M. The effect of omega-3 fatty acids supplementation on social and behavioral disorders of children with autism: a randomized clinical trial. Pediatr Endocrinol Diabetes Metab. 2021;27(1):12-18. doi: 10.5114/pedm.2020.101806. PMID 33599431
- [Background] Yehuda S, Rabinovitz-Shenkar S, Carasso RL. Effects of essential fatty acids in iron deficient and sleep-disturbed attention deficit hyperactivity disorder (ADHD) children. Eur J Clin Nutr. 2011 Oct;65(10):1167-9. doi: 10.1038/ejcn.2011.80. Epub 2011 May 18. PMID 21587279
- [Background] Grosso G, Micek A, Marventano S, Castellano S, Mistretta A, Pajak A, Galvano F. Dietary n-3 PUFA, fish consumption and depression: A systematic review and meta-analysis of observational studies. J Affect Disord. 2016 Nov 15;205:269-281. doi: 10.1016/j.jad.2016.08.011. Epub 2016 Aug 16. PMID 27544316
- [Background] Nemets H, Nemets B, Apter A, Bracha Z, Belmaker RH. Omega-3 treatment of childhood depression: a controlled, double-blind pilot study. Am J Psychiatry. 2006 Jun;163(6):1098-100. doi: 10.1176/ajp.2006.163.6.1098. PMID 16741212
- [Background] Minns LM, Kerling EH, Neely MR, Sullivan DK, Wampler JL, Harris CL, Berseth CL, Carlson SE. Toddler formula supplemented with docosahexaenoic acid (DHA) improves DHA status and respiratory health in a randomized, double-blind, controlled trial of US children less than 3 years of age. Prostaglandins Leukot Essent Fatty Acids. 2010 Apr-Jun;82(4-6):287-93. doi: 10.1016/j.plefa.2010.02.009. Epub 2010 Mar 5. PMID 20207123
- [Background] Czumaj A, Sledzinski T. Biological Role of Unsaturated Fatty Acid Desaturases in Health and Disease. Nutrients. 2020 Jan 29;12(2):356. doi: 10.3390/nu12020356. PMID 32013225
- [Background] Muc M, Kreiner-Moller E, Larsen JM, Birch S, Brix S, Bisgaard H, Lauritzen L. Maternal fatty acid desaturase genotype correlates with infant immune responses at 6 months. Br J Nutr. 2015 Sep 28;114(6):891-8. doi: 10.1017/S0007114515002561. Epub 2015 Aug 18. PMID 26283408
- [Background] Bazinet RP, Laye S. Polyunsaturated fatty acids and their metabolites in brain function and disease. Nat Rev Neurosci. 2014 Dec;15(12):771-85. doi: 10.1038/nrn3820. Epub 2014 Nov 12. PMID 25387473
- [Background] Madore C, Leyrolle Q, Lacabanne C, Benmamar-Badel A, Joffre C, Nadjar A, Laye S. Neuroinflammation in Autism: Plausible Role of Maternal Inflammation, Dietary Omega 3, and Microbiota. Neural Plast. 2016;2016:3597209. doi: 10.1155/2016/3597209. Epub 2016 Oct 20. PMID 27840741
- [Background] AlAmmar WA, Albeesh FH, Ibrahim LM, Algindan YY, Yamani LZ, Khattab RY. Effect of omega-3 fatty acids and fish oil supplementation on multiple sclerosis: a systematic review. Nutr Neurosci. 2021 Jul;24(7):569-579. doi: 10.1080/1028415X.2019.1659560. Epub 2019 Aug 28. PMID 31462182
- [Background] Wei BZ, Li L, Dong CW, Tan CC; Alzheimer's Disease Neuroimaging Initiative; Xu W. The Relationship of Omega-3 Fatty Acids with Dementia and Cognitive Decline: Evidence from Prospective Cohort Studies of Supplementation, Dietary Intake, and Blood Markers. Am J Clin Nutr. 2023 Jun;117(6):1096-1109. doi: 10.1016/j.ajcnut.2023.04.001. Epub 2023 Apr 5. PMID 37028557
- [Background] Riediger ND, Othman RA, Suh M, Moghadasian MH. A systemic review of the roles of n-3 fatty acids in health and disease. J Am Diet Assoc. 2009 Apr;109(4):668-79. doi: 10.1016/j.jada.2008.12.022. PMID 19328262
- [Background] Dou Y, Wang Y, Chen Z, Yu X, Ma D. Effect of n-3 polyunsaturated fatty acid on bone health: A systematic review and meta-analysis of randomized controlled trials. Food Sci Nutr. 2021 Nov 29;10(1):145-154. doi: 10.1002/fsn3.2655. eCollection 2022 Jan. PMID 35035917
- [Background] Goldberg RJ, Katz J. A meta-analysis of the analgesic effects of omega-3 polyunsaturated fatty acid supplementation for inflammatory joint pain. Pain. 2007 May;129(1-2):210-23. doi: 10.1016/j.pain.2007.01.020. Epub 2007 Mar 1. PMID 17335973
- [Background] Liput KP, Lepczynski A, Ogluszka M, Nawrocka A, Polawska E, Grzesiak A, Slaska B, Pareek CS, Czarnik U, Pierzchala M. Effects of Dietary n-3 and n-6 Polyunsaturated Fatty Acids in Inflammation and Cancerogenesis. Int J Mol Sci. 2021 Jun 28;22(13):6965. doi: 10.3390/ijms22136965. PMID 34203461
- [Background] Sugawara E, Nikaido H. Properties of AdeABC and AdeIJK efflux systems of Acinetobacter baumannii compared with those of the AcrAB-TolC system of Escherichia coli. Antimicrob Agents Chemother. 2014 Dec;58(12):7250-7. doi: 10.1128/AAC.03728-14. Epub 2014 Sep 22. PMID 25246403
- [Background] Nienaber A, Ozturk M, Dolman R, Blaauw R, Zandberg LL, van Rensburg S, Britz M, Hayford FEA, Brombacher F, Loots DT, Smuts CM, Parihar SP, Malan L. n-3 long-chain PUFA promote antibacterial and inflammation-resolving effects in Mycobacterium tuberculosis-infected C3HeB/FeJ mice, dependent on fatty acid status. Br J Nutr. 2022 Feb 14;127(3):384-397. doi: 10.1017/S0007114521001124. Epub 2021 Apr 5. PMID 33814018
- [Background] Spooner MH, Jump DB. Omega-3 fatty acids and nonalcoholic fatty liver disease in adults and children: where do we stand? Curr Opin Clin Nutr Metab Care. 2019 Mar;22(2):103-110. doi: 10.1097/MCO.0000000000000539. PMID 30601174
- [Background] Siriwardhana N, Kalupahana NS, Moustaid-Moussa N. Health benefits of n-3 polyunsaturated fatty acids: eicosapentaenoic acid and docosahexaenoic acid. Adv Food Nutr Res. 2012;65:211-22. doi: 10.1016/B978-0-12-416003-3.00013-5. PMID 22361189
- [Background] Chalon S. Omega-3 fatty acids and monoamine neurotransmission. Prostaglandins Leukot Essent Fatty Acids. 2006 Oct-Nov;75(4-5):259-69. doi: 10.1016/j.plefa.2006.07.005. Epub 2006 Sep 11. PMID 16963244
- [Background] Nordoy A, Marchioli R, Arnesen H, Videbaek J. n-3 polyunsaturated fatty acids and cardiovascular diseases. Lipids. 2001;36 Suppl:S127-9. doi: 10.1007/s11745-001-0695-7. PMID 11837986
- [Background] Landymore RW, Manku MS, Tan M, MacAulay MA, Sheridan B. Effects of low-dose marine oils on intimal hyperplasia in autologous vein grafts. J Thorac Cardiovasc Surg. 1989 Nov;98(5 Pt 1):788-91. PMID 2554068
- [Background] Pradelli L, Mayer K, Muscaritoli M, Heller AR. n-3 fatty acid-enriched parenteral nutrition regimens in elective surgical and ICU patients: a meta-analysis. Crit Care. 2012 Oct 4;16(5):R184. doi: 10.1186/cc11668. PMID 23036226
- [Background] Abeywardena MY, Head RJ. Longchain n-3 polyunsaturated fatty acids and blood vessel function. Cardiovasc Res. 2001 Dec;52(3):361-71. doi: 10.1016/s0008-6363(01)00406-0. PMID 11738053
- [Background] Jahangiri A, Leifert WR, Patten GS, McMurchie EJ. Termination of asynchronous contractile activity in rat atrial myocytes by n-3 polyunsaturated fatty acids. Mol Cell Biochem. 2000 Mar;206(1-2):33-41. doi: 10.1023/a:1007025007403. PMID 10839192
- [Background] Mozaffarian D, Psaty BM, Rimm EB, Lemaitre RN, Burke GL, Lyles MF, Lefkowitz D, Siscovick DS. Fish intake and risk of incident atrial fibrillation. Circulation. 2004 Jul 27;110(4):368-73. doi: 10.1161/01.CIR.0000138154.00779.A5. Epub 2004 Jul 19. PMID 15262826
- [Background] Thies F, Garry JM, Yaqoob P, Rerkasem K, Williams J, Shearman CP, Gallagher PJ, Calder PC, Grimble RF. Association of n-3 polyunsaturated fatty acids with stability of atherosclerotic plaques: a randomised controlled trial. Lancet. 2003 Feb 8;361(9356):477-85. doi: 10.1016/S0140-6736(03)12468-3. PMID 12583947
- [Background] Mozaffarian D. Fish, n-3 fatty acids, and cardiovascular haemodynamics. J Cardiovasc Med (Hagerstown). 2007 Sep;8 Suppl 1:S23-6. doi: 10.2459/01.JCM.0000289279.95427.e2. PMID 17876193
- [Background] Saremi A, Arora R. The utility of omega-3 fatty acids in cardiovascular disease. Am J Ther. 2009 Sep-Oct;16(5):421-36. doi: 10.1097/MJT.0b013e3180a5f0bb. PMID 19092647
- [Background] Russo GL. Dietary n-6 and n-3 polyunsaturated fatty acids: from biochemistry to clinical implications in cardiovascular prevention. Biochem Pharmacol. 2009 Mar 15;77(6):937-46. doi: 10.1016/j.bcp.2008.10.020. Epub 2008 Oct 28. PMID 19022225
- [Background] Mori TA, Burke V, Puddey IB, Watts GF, O'Neal DN, Best JD, Beilin LJ. Purified eicosapentaenoic and docosahexaenoic acids have differential effects on serum lipids and lipoproteins, LDL particle size, glucose, and insulin in mildly hyperlipidemic men. Am J Clin Nutr. 2000 May;71(5):1085-94. doi: 10.1093/ajcn/71.5.1085. PMID 10799369
- [Background] Kalstad AA, Myhre PL, Laake K, Tveit SH, Schmidt EB, Smith P, Nilsen DWT, Tveit A, Fagerland MW, Solheim S, Seljeflot I, Arnesen H; OMEMI Investigators. Effects of n-3 Fatty Acid Supplements in Elderly Patients After Myocardial Infarction: A Randomized, Controlled Trial. Circulation. 2021 Feb 9;143(6):528-539. doi: 10.1161/CIRCULATIONAHA.120.052209. Epub 2020 Nov 15. PMID 33191772
- [Background] Albert CM, Campos H, Stampfer MJ, Ridker PM, Manson JE, Willett WC, Ma J. Blood levels of long-chain n-3 fatty acids and the risk of sudden death. N Engl J Med. 2002 Apr 11;346(15):1113-8. doi: 10.1056/NEJMoa012918. PMID 11948270
- [Background] Siscovick DS, Raghunathan T, King I, Weinmann S, Bovbjerg VE, Kushi L, Cobb LA, Copass MK, Psaty BM, Lemaitre R, Retzlaff B, Knopp RH. Dietary intake of long-chain n-3 polyunsaturated fatty acids and the risk of primary cardiac arrest. Am J Clin Nutr. 2000 Jan;71(1 Suppl):208S-12S. doi: 10.1093/ajcn/71.1.208S. PMID 10617973
- [Background] Lemaitre RN, King IB, Mozaffarian D, Kuller LH, Tracy RP, Siscovick DS. n-3 Polyunsaturated fatty acids, fatal ischemic heart disease, and nonfatal myocardial infarction in older adults: the Cardiovascular Health Study. Am J Clin Nutr. 2003 Feb;77(2):319-25. doi: 10.1093/ajcn/77.2.319. PMID 12540389
- [Background] Shahidi F, Ambigaipalan P. Omega-3 Polyunsaturated Fatty Acids and Their Health Benefits. Annu Rev Food Sci Technol. 2018 Mar 25;9:345-381. doi: 10.1146/annurev-food-111317-095850. PMID 29350557
- [Background] Calder PC, Yaqoob P. Omega-3 polyunsaturated fatty acids and human health outcomes. Biofactors. 2009 May-Jun;35(3):266-72. doi: 10.1002/biof.42. PMID 19391122
- [Background] Bhatt DL, Steg PG, Brinton EA, Jacobson TA, Miller M, Tardif JC, Ketchum SB, Doyle RT Jr, Murphy SA, Soni PN, Braeckman RA, Juliano RA, Ballantyne CM; REDUCE-IT Investigators. Rationale and design of REDUCE-IT: Reduction of Cardiovascular Events with Icosapent Ethyl-Intervention Trial. Clin Cardiol. 2017 Mar;40(3):138-148. doi: 10.1002/clc.22692. Epub 2017 Mar 15. PMID 28294373
- [Background] AHA; ACC; National Heart, Lung, and Blood Institute; Smith SC Jr, Allen J, Blair SN, Bonow RO, Brass LM, Fonarow GC, Grundy SM, Hiratzka L, Jones D, Krumholz HM, Mosca L, Pearson T, Pfeffer MA, Taubert KA. AHA/ACC guidelines for secondary prevention for patients with coronary and other atherosclerotic vascular disease: 2006 update endorsed by the National Heart, Lung, and Blood Institute. J Am Coll Cardiol. 2006 May 16;47(10):2130-9. doi: 10.1016/j.jacc.2006.04.026. No abstract available. PMID 16697342
- [Background] Lomivorotov VV, Efremov SM, Pokushalov EA, Romanov AB, Ponomarev DN, Cherniavsky AM, Shilova AN, Karaskov AM, Lomivorotov VN. Randomized trial of fish oil infusion to prevent atrial fibrillation after cardiac surgery: data from an implantable continuous cardiac monitor. J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1278-84. doi: 10.1053/j.jvca.2014.02.019. Epub 2014 Jul 11. PMID 25027101
- [Background] Mayo Clinic Staff. Fish oil. Mayo Clinic Press. August 10, 2023. Accessed October 23, 2024. https://www.mayoclinic.org/drugs-supplements-fish-oil/art-20364810
- [Background] Souza PR, Marques RM, Gomez EA, Colas RA, De Matteis R, Zak A, Patel M, Collier DJ, Dalli J. Enriched Marine Oil Supplements Increase Peripheral Blood Specialized Pro-Resolving Mediators Concentrations and Reprogram Host Immune Responses: A Randomized Double-Blind Placebo-Controlled Study. Circ Res. 2020 Jan 3;126(1):75-90. doi: 10.1161/CIRCRESAHA.119.315506. Epub 2019 Dec 12. PMID 31829100
- [Background] Simopoulos AP. The importance of the ratio of omega-6/omega-3 essential fatty acids. Biomed Pharmacother. 2002 Oct;56(8):365-79. doi: 10.1016/s0753-3322(02)00253-6. PMID 12442909
- [Background] Djuricic I, Calder PC. Pros and Cons of Long-Chain Omega-3 Polyunsaturated Fatty Acids in Cardiovascular Health. Annu Rev Pharmacol Toxicol. 2023 Jan 20;63:383-406. doi: 10.1146/annurev-pharmtox-051921-090208. PMID 36662586
- [Background] von Schacky C, Fischer S, Weber PC. Long-term effects of dietary marine omega-3 fatty acids upon plasma and cellular lipids, platelet function, and eicosanoid formation in humans. J Clin Invest. 1985 Oct;76(4):1626-31. doi: 10.1172/JCI112147. PMID 2997286
- [Background] Biasi E. The effects of dietary choline. Neurosci Bull. 2011 Oct;27(5):330-42. doi: 10.1007/s12264-011-1523-5. PMID 21934729
- [Background] Zhang B, Zhen Y, Tao A, Bao Z, Zhang G. Polyunsaturated fatty acids for the prevention of atrial fibrillation after cardiac surgery: an updated meta-analysis of randomized controlled trials. J Cardiol. 2014 Jan;63(1):53-9. doi: 10.1016/j.jjcc.2013.06.014. Epub 2013 Aug 1. PMID 23911138
- [Background] Langlois PL, Hardy G, Manzanares W. Omega-3 polyunsaturated fatty acids in cardiac surgery patients: An updated systematic review and meta-analysis. Clin Nutr. 2017 Jun;36(3):737-746. doi: 10.1016/j.clnu.2016.05.013. Epub 2016 May 27. PMID 27293143
- [Background] Veljovic M, Mihajlovic I, Subota V, Antunovic M, Jevdjic J, Udovicic I, Popadic A, Vulovic T. Effect of pretreatment with omega-3 polyunsaturated fatty acids (PUfas) on hematological parameters and platelets aggregation in patients during elective coronary artery bypass grafting. Vojnosanit Pregl. 2013 Apr;70(4):396-402. doi: 10.2298/vsp1304396v. PMID 23700945
- [Background] Harker LA, Kelly AB, Hanson SR, Krupski W, Bass A, Osterud B, FitzGerald GA, Goodnight SH, Connor WE. Interruption of vascular thrombus formation and vascular lesion formation by dietary n-3 fatty acids in fish oil in nonhuman primates. Circulation. 1993 Mar;87(3):1017-29. doi: 10.1161/01.cir.87.3.1017. PMID 8443878
- [Background] Veljovic M, Popadic A, Vukic Z, Ilic R, Trifunovic Z, Antunovic M, Mandaric V, Tisma S, Markovic Z. Myocardial protection during elective coronary artery bypasses grafting by pretreatment with omega-3 polyunsaturated fatty acids. Vojnosanit Pregl. 2013 May;70(5):484-92. doi: 10.2298/vsp1305484v. PMID 23789288
- [Background] Stanger O, Aigner I, Schimetta W, Wonisch W. Antioxidant supplementation attenuates oxidative stress in patients undergoing coronary artery bypass graft surgery. Tohoku J Exp Med. 2014 Feb;232(2):145-54. doi: 10.1620/tjem.232.145. PMID 24573122
- [Background] Gholami M, Najafizadeh H, Teimouri H, Ardalan A, Pooria A, Tarrahi MJ. The combined effect of vitamin C and omega-3 polyunsaturated fatty acids on fatigue following coronary artery bypass graft surgery: a triple-blind clinical trial. J Complement Integr Med. 2019 Aug 21;16(4):/j/jcim.2019.16.issue-4/jcim-2018-0113/jcim-2018-0113.xml. doi: 10.1515/jcim-2018-0113. PMID 31433781
- [Background] Feguri GR, Lima PRL, Franco AC, Cruz FRH, Borges DC, Toledo LR, Segri NJ, Aguilar-Nascimento JE. Benefits of Fasting Abbreviation with Carbohydrates and Omega-3 Infusion During CABG: a Double-Blind Controlled Randomized Trial. Braz J Cardiovasc Surg. 2019 Mar-Apr;34(2):125-135. doi: 10.21470/1678-9741-2018-0336. PMID 30916121
- [Background] Mariscalco G, Sarzi Braga S, Banach M, Borsani P, Bruno VD, Napoleone M, Vitale C, Piffaretti G, Pedretti RF, Sala A. Preoperative n-3 polyunsatured fatty acids are associated with a decrease in the incidence of early atrial fibrillation following cardiac surgery. Angiology. 2010 Oct;61(7):643-50. doi: 10.1177/0003319710370962. Epub 2010 Jun 7. PMID 20529975
- [Background] Hagenfeldt L. Renal excretion of free fatty acids. Clin Chim Acta. 1971 May;32(3):471-4. doi: 10.1016/0009-8981(71)90450-5. No abstract available. PMID 5096958
- [Background] Dyerberg J, Madsen P, Moller JM, Aardestrup I, Schmidt EB. Bioavailability of marine n-3 fatty acid formulations. Prostaglandins Leukot Essent Fatty Acids. 2010 Sep;83(3):137-41. doi: 10.1016/j.plefa.2010.06.007. PMID 20638827
- [Background] Nelson GJ, Ackman RG. Absorption and transport of fat in mammals with emphasis on n-3 polyunsaturated fatty acids. Lipids. 1988 Nov;23(11):1005-14. doi: 10.1007/BF02535644. PMID 3070250
- [Background] Corsetto PA, Cremona A, Montorfano G, Jovenitti IE, Orsini F, Arosio P, Rizzo AM. Chemical-physical changes in cell membrane microdomains of breast cancer cells after omega-3 PUFA incorporation. Cell Biochem Biophys. 2012 Sep;64(1):45-59. doi: 10.1007/s12013-012-9365-y. PMID 22622660
- [Background] Jump DB. The biochemistry of n-3 polyunsaturated fatty acids. J Biol Chem. 2002 Mar 15;277(11):8755-8. doi: 10.1074/jbc.R100062200. Epub 2001 Dec 17. No abstract available. PMID 11748246
- [Background] Valentine RC, Valentine DL. Omega-3 fatty acids in cellular membranes: a unified concept. Prog Lipid Res. 2004 Sep;43(5):383-402. doi: 10.1016/j.plipres.2004.05.004. PMID 15458813
- [Background] Mason RP, Libby P, Bhatt DL. Emerging Mechanisms of Cardiovascular Protection for the Omega-3 Fatty Acid Eicosapentaenoic Acid. Arterioscler Thromb Vasc Biol. 2020 May;40(5):1135-1147. doi: 10.1161/ATVBAHA.119.313286. Epub 2020 Mar 26. PMID 32212849
- [Background] Masson S, Wu JH, Simon C, Barlera S, Marchioli R, Mariani J, Macchia A, Lombardi F, Vago T, Aleksova A, Dreas L, Favaloro RR, Hershson AR, Puskas JD, Dozza L, Silletta MG, Tognoni G, Mozaffarian D, Latini R; OPERA Investigators. Circulating cardiac biomarkers and postoperative atrial fibrillation in the OPERA trial. Eur J Clin Invest. 2015 Feb;45(2):170-8. doi: 10.1111/eci.12393. Epub 2015 Jan 7. PMID 25510286
- [Background] Vasheghani Farahani A, Yousefi Azar A, Goodarzynejad HR, Khorrami E, Hosseinzadeh-Attar MJ, Oshnouei S, Alizadeh Ghavidel A, Golfeshan E, Ghourban Pour F. Fish oil supplementation for primary prevention of atrial fibrillation after coronary artery bypass graft surgery: A randomized clinical trial. Int J Surg. 2017 Jun;42:41-48. doi: 10.1016/j.ijsu.2017.04.025. Epub 2017 Apr 15. PMID 28419884
- [Background] Sorice M, Tritto FP, Sordelli C, Gregorio R, Piazza L. N-3 polyunsaturated fatty acids reduces post-operative atrial fibrillation incidence in patients undergoing "on-pump" coronary artery bypass graft surgery. Monaldi Arch Chest Dis. 2011 Jun;76(2):93-8. doi: 10.4081/monaldi.2011.196. PMID 22128614
- [Background] Calo L, Bianconi L, Colivicchi F, Lamberti F, Loricchio ML, de Ruvo E, Meo A, Pandozi C, Staibano M, Santini M. N-3 Fatty acids for the prevention of atrial fibrillation after coronary artery bypass surgery: a randomized, controlled trial. J Am Coll Cardiol. 2005 May 17;45(10):1723-8. doi: 10.1016/j.jacc.2005.02.079. PMID 15893193
- [Background] Charman A, Muriithi EW, Milne E, Wheatley DJ, Armstrong RA, Belcher PR. Fish oil before cardiac surgery: neutrophil activation is unaffected but myocardial damage is moderated. Prostaglandins Leukot Essent Fatty Acids. 2005 Apr;72(4):257-65. doi: 10.1016/j.plefa.2004.11.007. PMID 15763437
- [Background] Benedetto U, Melina G, di Bartolomeo R, Angeloni E, Sansone D, Falaschi G, Capuano F, Comito C, Roscitano A, Sinatra R. n-3 polyunsaturated fatty acids after coronary artery bypass grafting. Ann Thorac Surg. 2011 Apr;91(4):1169-75. doi: 10.1016/j.athoracsur.2010.11.068. PMID 21440140
- [Background] Castillo R, Rodrigo R, Perez F, Cereceda M, Asenjo R, Zamorano J, Navarrete R, Villalabeitia E, Sanz J, Baeza C, Aguayo R. Antioxidant therapy reduces oxidative and inflammatory tissue damage in patients subjected to cardiac surgery with extracorporeal circulation. Basic Clin Pharmacol Toxicol. 2011 Apr;108(4):256-62. doi: 10.1111/j.1742-7843.2010.00651.x. Epub 2010 Dec 8. PMID 21138533
- [Background] Rodrigo R, Korantzopoulos P, Cereceda M, Asenjo R, Zamorano J, Villalabeitia E, Baeza C, Aguayo R, Castillo R, Carrasco R, Gormaz JG. A randomized controlled trial to prevent post-operative atrial fibrillation by antioxidant reinforcement. J Am Coll Cardiol. 2013 Oct 15;62(16):1457-65. doi: 10.1016/j.jacc.2013.07.014. Epub 2013 Jul 31. PMID 23916928
- [Background] Rodrigo R, Gutierrez R, Fernandez R, Guzman P. Ageing improves the antioxidant response against postoperative atrial fibrillation: a randomized controlled trial. Interact Cardiovasc Thorac Surg. 2012 Aug;15(2):209-14. doi: 10.1093/icvts/ivs154. Epub 2012 May 4. PMID 22561296
- [Background] National Institute of Health. Omega-3 fatty acids fact sheet for health professionals. NIH. 2023. https://ods.od.nih.gov/factsheets/Omega3FattyAcids-HealthProfessional/
- [Background] Skuladottir GV, Heidarsdottir R, Arnar DO, Torfason B, Edvardsson V, Gottskalksson G, Palsson R, Indridason OS. Plasma n-3 and n-6 fatty acids and the incidence of atrial fibrillation following coronary artery bypass graft surgery. Eur J Clin Invest. 2011 Sep;41(9):995-1003. doi: 10.1111/j.1365-2362.2011.02497.x. Epub 2011 Mar 17. PMID 21413975
- [Background] Akintoye E, Sethi P, Harris WS, Thompson PA, Marchioli R, Tavazzi L, Latini R, Pretorius M, Brown NJ, Libby P, Mozaffarian D. Fish Oil and Perioperative Bleeding. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e004584. doi: 10.1161/CIRCOUTCOMES.118.004584. PMID 30571332
- [Background] Berger MM, Delodder F, Liaudet L, Tozzi P, Schlaepfer J, Chiolero RL, Tappy L. Three short perioperative infusions of n-3 PUFAs reduce systemic inflammation induced by cardiopulmonary bypass surgery: a randomized controlled trial. Am J Clin Nutr. 2013 Feb;97(2):246-54. doi: 10.3945/ajcn.112.046573. Epub 2012 Dec 26. PMID 23269816
- [Background] Eritsland J, Arnesen H, Seljeflot I, Kierulf P. Long-term effects of n-3 polyunsaturated fatty acids on haemostatic variables and bleeding episodes in patients with coronary artery disease. Blood Coagul Fibrinolysis. 1995 Feb;6(1):17-22. doi: 10.1097/00001721-199502000-00003. PMID 7795149
- [Background] Gu J, Lundbye-Christensen S, Eschen RB, Andreasen A, Andreasen JJ. Marine n-3 fatty acids are incorporated into atrial tissue but do not correlate with postoperative atrial fibrillation in cardiac surgery. Vascul Pharmacol. 2016 Dec;87:70-75. doi: 10.1016/j.vph.2016.11.004. Epub 2016 Nov 17. PMID 27867031
- [Background] Mozaffarian D, Marchioli R, Macchia A, Silletta MG, Ferrazzi P, Gardner TJ, Latini R, Libby P, Lombardi F, O'Gara PT, Page RL, Tavazzi L, Tognoni G; OPERA Investigators. Fish oil and postoperative atrial fibrillation: the Omega-3 Fatty Acids for Prevention of Post-operative Atrial Fibrillation (OPERA) randomized trial. JAMA. 2012 Nov 21;308(19):2001-11. doi: 10.1001/jama.2012.28733. PMID 23128104
- [Background] Jackson JC, Mozaffarian D, Graves AJ, Brown NJ, Marchioli R, Kiehl AL, Ely EW. Fish Oil Supplementation Does Not Affect Cognitive Outcomes in Cardiac Surgery Patients in the Omega-3 Fatty Acids for Prevention of Post-Operative Atrial Fibrillation (OPERA) Trial. J Nutr. 2018 Mar 1;148(3):472-479. doi: 10.1093/jn/nxx002. PMID 29546292
- [Background] Sandesara CM, Chung MK, Van Wagoner DR, Barringer TA, Allen K, Ismail HM, Zimmerman B, Olshansky B. A Randomized, Placebo-Controlled Trial of Omega-3 Fatty Acids for Inhibition of Supraventricular Arrhythmias After Cardiac Surgery: The FISH Trial. J Am Heart Assoc. 2012 Jun;1(3):e000547. doi: 10.1161/JAHA.111.000547. Epub 2012 Jun 22. PMID 23130134
- [Background] Saravanan P, Bridgewater B, West AL, O'Neill SC, Calder PC, Davidson NC. Omega-3 fatty acid supplementation does not reduce risk of atrial fibrillation after coronary artery bypass surgery: a randomized, double-blind, placebo-controlled clinical trial. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):46-53. doi: 10.1161/CIRCEP.109.899633. Epub 2009 Dec 30. PMID 20042769
- [Background] Akintoye E, Wu JH, Hou T, Song X, Yang J, Hammock B, Mozaffarian D. Effect of fish oil on monoepoxides derived from fatty acids during cardiac surgery. J Lipid Res. 2016 Mar;57(3):492-8. doi: 10.1194/jlr.P062398. Epub 2016 Jan 9. PMID 26749073
- [Background] Farquharson AL, Metcalf RG, Sanders P, Stuklis R, Edwards JR, Gibson RA, Cleland LG, Sullivan TR, James MJ, Young GD. Effect of dietary fish oil on atrial fibrillation after cardiac surgery. Am J Cardiol. 2011 Sep 15;108(6):851-6. doi: 10.1016/j.amjcard.2011.04.036. Epub 2011 Jul 15. PMID 21762871
- [Background] Heidarsdottir R, Arnar DO, Skuladottir GV, Torfason B, Edvardsson V, Gottskalksson G, Palsson R, Indridason OS. Does treatment with n-3 polyunsaturated fatty acids prevent atrial fibrillation after open heart surgery? Europace. 2010 Mar;12(3):356-63. doi: 10.1093/europace/eup429. Epub 2010 Jan 7. PMID 20061328
- [Background] Eritsland J, Arnesen H, Gronseth K, Fjeld NB, Abdelnoor M. Effect of dietary supplementation with n-3 fatty acids on coronary artery bypass graft patency. Am J Cardiol. 1996 Jan 1;77(1):31-6. doi: 10.1016/s0002-9149(97)89130-8. PMID 8540453
- [Background] Andreassen AK, Hartmann A, Offstad J, Geiran O, Kvernebo K, Simonsen S. Hypertension prophylaxis with omega-3 fatty acids in heart transplant recipients. J Am Coll Cardiol. 1997 May;29(6):1324-31. doi: 10.1016/s0735-1097(97)82757-x. PMID 9137231
- [Background] Rubanenko OA, Shchukin YV, Limareva LV, et al. Omega-3 polyunsaturated fatty acids: the role in prevention of atrial fibrillation in patients with coronary artery disease after coronary artery bypass graft surgery. Ration Pharmacother Cardiol 2022;18:12-19.
- [Background] Kim HY. Analysis of variance (ANOVA) comparing means of more than two groups. Restor Dent Endod. 2014 Feb;39(1):74-7. doi: 10.5395/rde.2014.39.1.74. No abstract available. PMID 24516834
- [Background] Rosner BA. Fundamentals of Biostatistics. Thomson-Brooks/Cole; 2006.
- [Background] He Z, Yang L, Tian J, Yang K, Wu J, Yao Y. Efficacy and safety of omega-3 fatty acids for the prevention of atrial fibrillation: a meta-analysis. Can J Cardiol. 2013 Feb;29(2):196-203. doi: 10.1016/j.cjca.2012.03.019. Epub 2012 Jun 7. PMID 22681963
- [Background] Costanzo S, di Niro V, Di Castelnuovo A, Gianfagna F, Donati MB, de Gaetano G, Iacoviello L. Prevention of postoperative atrial fibrillation in open heart surgery patients by preoperative supplementation of n-3 polyunsaturated fatty acids: an updated meta-analysis. J Thorac Cardiovasc Surg. 2013 Oct;146(4):906-11. doi: 10.1016/j.jtcvs.2013.03.015. Epub 2013 Apr 12. PMID 23587470
- [Background] Takagi H, Umemoto T. Preoperative n-3 Polyunsatured fatty acids do not reduce postoperative atrial fibrillation in cardiac surgery. Angiology. 2011 Apr;62(3):276-7; author reply 278-9. doi: 10.1177/0003319710389021. No abstract available. PMID 21406425
- [Background] Rinninella E, Costantini L. Polyunsaturated Fatty Acids as Prebiotics: Innovation or Confirmation? Foods. 2022 Jan 6;11(2):146. doi: 10.3390/foods11020146. PMID 35053879
- [Background] Costantini L, Molinari R, Farinon B, Merendino N. Impact of Omega-3 Fatty Acids on the Gut Microbiota. Int J Mol Sci. 2017 Dec 7;18(12):2645. doi: 10.3390/ijms18122645. PMID 29215589
- [Background] Shaikh SR, Edidin M. Polyunsaturated fatty acids and membrane organization: elucidating mechanisms to balance immunotherapy and susceptibility to infection. Chem Phys Lipids. 2008 May;153(1):24-33. doi: 10.1016/j.chemphyslip.2008.02.008. Epub 2008 Feb 23. PMID 18346461
- [Background] Hughes DA, Pinder AC. N-3 polyunsaturated fatty acids modulate the expression of functionally associated molecules on human monocytes and inhibit antigen-presentation in vitro. Clin Exp Immunol. 1997 Dec;110(3):516-23. doi: 10.1046/j.1365-2249.1997.4351455.x. PMID 9409659
- [Background] Asimakopoulos G, Smith PL, Ratnatunga CP, Taylor KM. Lung injury and acute respiratory distress syndrome after cardiopulmonary bypass. Ann Thorac Surg. 1999 Sep;68(3):1107-15. doi: 10.1016/s0003-4975(99)00781-x. PMID 10510030
- [Background] Calder PC. Omega-3 polyunsaturated fatty acids and inflammatory processes: nutrition or pharmacology? Br J Clin Pharmacol. 2013 Mar;75(3):645-62. doi: 10.1111/j.1365-2125.2012.04374.x. PMID 22765297
- [Background] Erkkila AT, Matthan NR, Herrington DM, Lichtenstein AH. Higher plasma docosahexaenoic acid is associated with reduced progression of coronary atherosclerosis in women with CAD. J Lipid Res. 2006 Dec;47(12):2814-9. doi: 10.1194/jlr.P600005-JLR200. Epub 2006 Sep 18. PMID 16983146
- [Background] Mozaffarian D, Rimm EB. Fish intake, contaminants, and human health: evaluating the risks and the benefits. JAMA. 2006 Oct 18;296(15):1885-99. doi: 10.1001/jama.296.15.1885. PMID 17047219
- [Background] Jump DB, Depner CM, Tripathy S. Omega-3 fatty acid supplementation and cardiovascular disease. J Lipid Res. 2012 Dec;53(12):2525-45. doi: 10.1194/jlr.R027904. Epub 2012 Aug 17. PMID 22904344
- [Background] Harris WS, Miller M, Tighe AP, Davidson MH, Schaefer EJ. Omega-3 fatty acids and coronary heart disease risk: clinical and mechanistic perspectives. Atherosclerosis. 2008 Mar;197(1):12-24. doi: 10.1016/j.atherosclerosis.2007.11.008. Epub 2007 Dec 26. PMID 18160071
- [Background] Jung UJ, Torrejon C, Tighe AP, Deckelbaum RJ. n-3 Fatty acids and cardiovascular disease: mechanisms underlying beneficial effects. Am J Clin Nutr. 2008 Jun;87(6):2003S-9S. doi: 10.1093/ajcn/87.6.2003S. PMID 18541602
- [Background] Watanabe Y, Tatsuno I. Omega-3 polyunsaturated fatty acids for cardiovascular diseases: present, past and future. Expert Rev Clin Pharmacol. 2017 Aug;10(8):865-873. doi: 10.1080/17512433.2017.1333902. Epub 2017 May 29. PMID 28531360
- [Background] Marchioli R, Barzi F, Bomba E, Chieffo C, Di Gregorio D, Di Mascio R, Franzosi MG, Geraci E, Levantesi G, Maggioni AP, Mantini L, Marfisi RM, Mastrogiuseppe G, Mininni N, Nicolosi GL, Santini M, Schweiger C, Tavazzi L, Tognoni G, Tucci C, Valagussa F; GISSI-Prevenzione Investigators. Early protection against sudden death by n-3 polyunsaturated fatty acids after myocardial infarction: time-course analysis of the results of the Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto Miocardico (GISSI)-Prevenzione. Circulation. 2002 Apr 23;105(16):1897-903. doi: 10.1161/01.cir.0000014682.14181.f2. PMID 11997274
- [Background] Leaf A. The electrophysiological basis for the antiarrhythmic actions of polyunsaturated fatty acids. Eur Heart J Suppl 2001;3:98-105.
- [Background] Leaf A, Albert CM, Josephson M, Steinhaus D, Kluger J, Kang JX, Cox B, Zhang H, Schoenfeld D; Fatty Acid Antiarrhythmia Trial Investigators. Prevention of fatal arrhythmias in high-risk subjects by fish oil n-3 fatty acid intake. Circulation. 2005 Nov 1;112(18):2762-8. doi: 10.1161/CIRCULATIONAHA.105.549527. PMID 16267249
- [Background] Leaf A, Kang JX, Xiao YF, Billman GE. Clinical prevention of sudden cardiac death by n-3 polyunsaturated fatty acids and mechanism of prevention of arrhythmias by n-3 fish oils. Circulation. 2003 Jun 3;107(21):2646-52. doi: 10.1161/01.CIR.0000069566.78305.33. No abstract available. PMID 12782616
- [Background] Merendino N, Costantini L, Manzi L, Molinari R, D'Eliseo D, Velotti F. Dietary omega -3 polyunsaturated fatty acid DHA: a potential adjuvant in the treatment of cancer. Biomed Res Int. 2013;2013:310186. doi: 10.1155/2013/310186. Epub 2013 May 23. PMID 23762838
- [Background] Arnold LE, Young AS, Belury MA, Cole RM, Gracious B, Seidenfeld AM, Wolfson H, Fristad MA. Omega-3 Fatty Acid Plasma Levels Before and After Supplementation: Correlations with Mood and Clinical Outcomes in the Omega-3 and Therapy Studies. J Child Adolesc Psychopharmacol. 2017 Apr;27(3):223-233. doi: 10.1089/cap.2016.0123. Epub 2017 Feb 3. PMID 28157380
- [Background] Calder PC. Polyunsaturated fatty acids, inflammation, and immunity. Lipids. 2001 Sep;36(9):1007-24. doi: 10.1007/s11745-001-0812-7. PMID 11724453
- [Background] Miles EA, Calder PC. Influence of marine n-3 polyunsaturated fatty acids on immune function and a systematic review of their effects on clinical outcomes in rheumatoid arthritis. Br J Nutr. 2012 Jun;107 Suppl 2:S171-84. doi: 10.1017/S0007114512001560. PMID 22591891
- [Background] Calder PC. n-3 Fatty acids and cardiovascular disease: evidence explained and mechanisms explored. Clin Sci (Lond). 2004 Jul;107(1):1-11. doi: 10.1042/CS20040119. PMID 15132735
- [Background] Zarate R, El Jaber-Vazdekis N, Tejera N, Perez JA, Rodriguez C. Significance of long chain polyunsaturated fatty acids in human health. Clin Transl Med. 2017 Dec;6(1):25. doi: 10.1186/s40169-017-0153-6. Epub 2017 Jul 27. PMID 28752333
- [Background] Yokoyama M, Origasa H, Matsuzaki M, Matsuzawa Y, Saito Y, Ishikawa Y, Oikawa S, Sasaki J, Hishida H, Itakura H, Kita T, Kitabatake A, Nakaya N, Sakata T, Shimada K, Shirato K; Japan EPA lipid intervention study (JELIS) Investigators. Effects of eicosapentaenoic acid on major coronary events in hypercholesterolaemic patients (JELIS): a randomised open-label, blinded endpoint analysis. Lancet. 2007 Mar 31;369(9567):1090-8. doi: 10.1016/S0140-6736(07)60527-3. PMID 17398308
- [Background] Burr ML, Fehily AM, Gilbert JF, Rogers S, Holliday RM, Sweetnam PM, Elwood PC, Deadman NM. Effects of changes in fat, fish, and fibre intakes on death and myocardial reinfarction: diet and reinfarction trial (DART). Lancet. 1989 Sep 30;2(8666):757-61. doi: 10.1016/s0140-6736(89)90828-3. PMID 2571009
- [Background] Nilsen DW, Albrektsen G, Landmark K, Moen S, Aarsland T, Woie L. Effects of a high-dose concentrate of n-3 fatty acids or corn oil introduced early after an acute myocardial infarction on serum triacylglycerol and HDL cholesterol. Am J Clin Nutr. 2001 Jul;74(1):50-6. doi: 10.1093/ajcn/74.1.50. PMID 11451717
- [Background] Heidt MC, Vician M, Stracke SK, Stadlbauer T, Grebe MT, Boening A, Vogt PR, Erdogan A. Beneficial effects of intravenously administered N-3 fatty acids for the prevention of atrial fibrillation after coronary artery bypass surgery: a prospective randomized study. Thorac Cardiovasc Surg. 2009 Aug;57(5):276-80. doi: 10.1055/s-0029-1185301. Epub 2009 Jul 23. PMID 19629889
- [Background] Kris-Etherton PM, Harris WS, Appel LJ; American Heart Association. Nutrition Committee. Fish consumption, fish oil, omega-3 fatty acids, and cardiovascular disease. Circulation. 2002 Nov 19;106(21):2747-57. doi: 10.1161/01.cir.0000038493.65177.94. No abstract available. PMID 12438303
- [Background] Kris-Etherton PM, Griel AE, Psota TL, Gebauer SK, Zhang J, Etherton TD. Dietary stearic acid and risk of cardiovascular disease: intake, sources, digestion, and absorption. Lipids. 2005 Dec;40(12):1193-200. doi: 10.1007/s11745-005-1485-y. PMID 16477802
- [Background] Mozaffarian D, Wu JH. Omega-3 fatty acids and cardiovascular disease: effects on risk factors, molecular pathways, and clinical events. J Am Coll Cardiol. 2011 Nov 8;58(20):2047-67. doi: 10.1016/j.jacc.2011.06.063. PMID 22051327
- [Background] Hooper L, Thompson RL, Harrison RA, Summerbell CD, Moore H, Worthington HV, Durrington PN, Ness AR, Capps NE, Davey Smith G, Riemersma RA, Ebrahim SB. Omega 3 fatty acids for prevention and treatment of cardiovascular disease. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD003177. doi: 10.1002/14651858.CD003177.pub2. PMID 15495044
- [Background] Krupa KN, Fritz K, Parmar M. Omega-3 Fatty Acids. 2024 Feb 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK564314/ PMID 33231984
- [Background] Scientific Advisory Committee on Nutrition (SACN). Saturated fats and health. Published online 2019:443. https://www.gov.uk/government/publications/saturated-fats-and-health-sacn-report
- [Background] EFSA. Scientific opinion on dietary reference values for fats, including saturated fatty acids, polyunsaturated fatty acids, monounsaturated fatty acids, trans fatty acids, and cholesterol. EFSA J 2016;8:1-107.
- [Background] Cholewski M, Tomczykowa M, Tomczyk M. A Comprehensive Review of Chemistry, Sources and Bioavailability of Omega-3 Fatty Acids. Nutrients. 2018 Nov 4;10(11):1662. doi: 10.3390/nu10111662. PMID 30400360
- [Background] Brouwer IA. Fish, Omega-3 Fatty Acids and Heart Disease. Woodhead Publishing Limited; 2008. doi: 10.1533/9781845694586.2.165.
- [Background] Calder PC. Mechanisms of action of (n-3) fatty acids. J Nutr. 2012 Mar;142(3):592S-599S. doi: 10.3945/jn.111.155259. Epub 2012 Jan 25. PMID 22279140
- [Background] Padayatty SJ, Sun AY, Chen Q, Espey MG, Drisko J, Levine M. Vitamin C: intravenous use by complementary and alternative medicine practitioners and adverse effects. PLoS One. 2010 Jul 7;5(7):e11414. doi: 10.1371/journal.pone.0011414. PMID 20628650
- [Background] Levine M, Padayatty SJ, Espey MG. Vitamin C: a concentration-function approach yields pharmacology and therapeutic discoveries. Adv Nutr. 2011 Mar;2(2):78-88. doi: 10.3945/an.110.000109. Epub 2011 Mar 10. PMID 22332036
- [Background] Levine M, Conry-Cantilena C, Wang Y, Welch RW, Washko PW, Dhariwal KR, Park JB, Lazarev A, Graumlich JF, King J, Cantilena LR. Vitamin C pharmacokinetics in healthy volunteers: evidence for a recommended dietary allowance. Proc Natl Acad Sci U S A. 1996 Apr 16;93(8):3704-9. doi: 10.1073/pnas.93.8.3704. PMID 8623000
- [Background] Meier ML, Pierce KN. New therapies for the treatment of heart failure with preserved ejection fraction. Am J Health Syst Pharm. 2022 Aug 19;79(17):1424-1430. doi: 10.1093/ajhp/zxac129. PMID 35524990
- [Background] Solomon SD, Vaduganathan M, L Claggett B, Packer M, Zile M, Swedberg K, Rouleau J, A Pfeffer M, Desai A, Lund LH, Kober L, Anand I, Sweitzer N, Linssen G, Merkely B, Luis Arango J, Vinereanu D, Chen CH, Senni M, Sibulo A, Boytsov S, Shi V, Rizkala A, Lefkowitz M, McMurray JJV. Sacubitril/Valsartan Across the Spectrum of Ejection Fraction in Heart Failure. Circulation. 2020 Feb 4;141(5):352-361. doi: 10.1161/CIRCULATIONAHA.119.044586. Epub 2019 Nov 17. PMID 31736342
- [Background] Hornig B, Arakawa N, Kohler C, Drexler H. Vitamin C improves endothelial function of conduit arteries in patients with chronic heart failure. Circulation. 1998 Feb 3;97(4):363-8. doi: 10.1161/01.cir.97.4.363. PMID 9468210
- [Background] Qin F, Yan C, Patel R, Liu W, Dong E. Vitamins C and E attenuate apoptosis, beta-adrenergic receptor desensitization, and sarcoplasmic reticular Ca2+ ATPase downregulation after myocardial infarction. Free Radic Biol Med. 2006 May 15;40(10):1827-42. doi: 10.1016/j.freeradbiomed.2006.01.019. Epub 2006 Feb 8. PMID 16678021
- [Background] Shinke T, Shite J, Takaoka H, Hata K, Inoue N, Yoshikawa R, Matsumoto H, Masai H, Watanabe S, Ozawa T, Otake H, Matsumoto D, Hirata K, Yokoyama M. Vitamin C restores the contractile response to dobutamine and improves myocardial efficiency in patients with heart failure after anterior myocardial infarction. Am Heart J. 2007 Oct;154(4):645.e1-8. doi: 10.1016/j.ahj.2007.07.005. PMID 17892985
- [Background] Hemila H, Chalker E, de Man AME. Vitamin C May Improve Left Ventricular Ejection Fraction: A Meta-Analysis. Front Cardiovasc Med. 2022 Feb 25;9:789729. doi: 10.3389/fcvm.2022.789729. eCollection 2022. PMID 35282368
- [Background] Khan SA, Bhattacharjee S, Ghani MOA, Walden R, Chen QM. Vitamin C for Cardiac Protection during Percutaneous Coronary Intervention: A Systematic Review of Randomized Controlled Trials. Nutrients. 2020 Jul 23;12(8):2199. doi: 10.3390/nu12082199. PMID 32718091
- [Background] Valls N, Gormaz JG, Aguayo R, Gonzalez J, Brito R, Hasson D, Libuy M, Ramos C, Carrasco R, Prieto JC, Dussaillant G, Puentes A, Noriega V, Rodrigo R. Amelioration of persistent left ventricular function impairment through increased plasma ascorbate levels following myocardial infarction. Redox Rep. 2016 Mar;21(2):75-83. doi: 10.1179/1351000215Y.0000000018. Epub 2016 Feb 24. PMID 26066587
- [Background] Rodrigo R, Prieto JC, Aguayo R, Ramos C, Puentes A, Gajardo A, Panieri E, Rojas-Sole C, Lillo-Moya J, Saso L. Joint Cardioprotective Effect of Vitamin C and Other Antioxidants against Reperfusion Injury in Patients with Acute Myocardial Infarction Undergoing Percutaneous Coronary Intervention. Molecules. 2021 Sep 21;26(18):5702. doi: 10.3390/molecules26185702. PMID 34577176
- [Background] Malik A, Bagchi AK, Vinayak K, Akolkar G, Slezak J, Bello-Klein A, Jassal DS, Singal PK. Vitamin C: historical perspectives and heart failure. Heart Fail Rev. 2021 May;26(3):699-709. doi: 10.1007/s10741-020-10036-y. Epub 2020 Oct 8. PMID 33033908
- [Background] Keith M, Geranmayegan A, Sole MJ, Kurian R, Robinson A, Omran AS, Jeejeebhoy KN. Increased oxidative stress in patients with congestive heart failure. J Am Coll Cardiol. 1998 May;31(6):1352-6. doi: 10.1016/s0735-1097(98)00101-6. PMID 9581732
- [Background] de Lorgeril M, Salen P, Accominotti M, Cadau M, Steghens JP, Boucher F, de Leiris J. Dietary and blood antioxidants in patients with chronic heart failure. Insights into the potential importance of selenium in heart failure. Eur J Heart Fail. 2001 Dec;3(6):661-9. doi: 10.1016/s1388-9842(01)00179-9. PMID 11738217
- [Background] Munzel T, Camici GG, Maack C, Bonetti NR, Fuster V, Kovacic JC. Impact of Oxidative Stress on the Heart and Vasculature: Part 2 of a 3-Part Series. J Am Coll Cardiol. 2017 Jul 11;70(2):212-229. doi: 10.1016/j.jacc.2017.05.035. PMID 28683969
- [Background] Szyller J, Jagielski D, Bil-Lula I. Antioxidants in Arrhythmia Treatment-Still a Controversy? A Review of Selected Clinical and Laboratory Research. Antioxidants (Basel). 2022 Jun 2;11(6):1109. doi: 10.3390/antiox11061109. PMID 35740006
- [Background] Baker WL, Coleman CI. Meta-analysis of ascorbic acid for prevention of postoperative atrial fibrillation after cardiac surgery. Am J Health Syst Pharm. 2016 Dec 15;73(24):2056-2066. doi: 10.2146/ajhp160066. Epub 2016 Nov 2. PMID 27806938
- [Background] Korantzopoulos P, Kolettis T, Siogas K, Goudevenos J. Atrial fibrillation and electrical remodeling: the potential role of inflammation and oxidative stress. Med Sci Monit. 2003 Sep;9(9):RA225-9. PMID 12960937
- [Background] Hemila H, Suonsyrja T. Vitamin C for preventing atrial fibrillation in high risk patients: a systematic review and meta-analysis. BMC Cardiovasc Disord. 2017 Feb 1;17(1):49. doi: 10.1186/s12872-017-0478-5. PMID 28143406
- [Background] Sacks GS. Randomized, prospective trial of antioxidant supplementation in critically iii surgical patients. Nutr Clin Pract 2003;18:264.
- [Background] Emadi N, Nemati MH, Ghorbani M, Allahyari E. The Effect of High-Dose Vitamin C on Biochemical Markers of Myocardial Injury in Coronary Artery Bypass Surgery. Braz J Cardiovasc Surg. 2019 Dec 1;34(5):517-524. doi: 10.21470/1678-9741-2018-0312. PMID 31719005
- [Background] Frei B, Stocker R, England L, Ames BN. Ascorbate: the most effective antioxidant in human blood plasma. Adv Exp Med Biol. 1990;264:155-63. doi: 10.1007/978-1-4684-5730-8_24. PMID 2244489
- [Background] Frei B, England L, Ames BN. Ascorbate is an outstanding antioxidant in human blood plasma. Proc Natl Acad Sci U S A. 1989 Aug;86(16):6377-81. doi: 10.1073/pnas.86.16.6377. PMID 2762330
- [Background] Snezhkina AV, Kudryavtseva AV, Kardymon OL, Savvateeva MV, Melnikova NV, Krasnov GS, Dmitriev AA. ROS Generation and Antioxidant Defense Systems in Normal and Malignant Cells. Oxid Med Cell Longev. 2019 Aug 5;2019:6175804. doi: 10.1155/2019/6175804. eCollection 2019. PMID 31467634
- [Background] Landis RC, Brown JR, Fitzgerald D, Likosky DS, Shore-Lesserson L, Baker RA, Hammon JW. Attenuating the Systemic Inflammatory Response to Adult Cardiopulmonary Bypass: A Critical Review of the Evidence Base. J Extra Corpor Technol. 2014 Sep;46(3):197-211. PMID 26357785
- [Background] Giakoumidakis K, Baltopoulos GI, Charitos C, Patelarou E, Galanis P, Brokalaki H. Risk factors for prolonged stay in cardiac surgery intensive care units. Nurs Crit Care. 2011 Sep-Oct;16(5):243-51. doi: 10.1111/j.1478-5153.2010.00443.x. PMID 21824229
- [Background] Butler J, Rocker GM, Westaby S. Inflammatory response to cardiopulmonary bypass. Ann Thorac Surg. 1993 Feb;55(2):552-9. doi: 10.1016/0003-4975(93)91048-r. PMID 8431082
- [Background] Hall R. Identification of inflammatory mediators and their modulation by strategies for the management of the systemic inflammatory response during cardiac surgery. J Cardiothorac Vasc Anesth. 2013 Oct;27(5):983-1033. doi: 10.1053/j.jvca.2012.09.013. Epub 2012 Dec 29. No abstract available. PMID 23276596
- [Background] Langlois M, Duprez D, Delanghe J, De Buyzere M, Clement DL. Serum vitamin C concentration is low in peripheral arterial disease and is associated with inflammation and severity of atherosclerosis. Circulation. 2001 Apr 10;103(14):1863-8. doi: 10.1161/01.cir.103.14.1863. PMID 11294804
- [Background] Yokoyama T, Date C, Kokubo Y, Yoshiike N, Matsumura Y, Tanaka H. Serum vitamin C concentration was inversely associated with subsequent 20-year incidence of stroke in a Japanese rural community. The Shibata study. Stroke. 2000 Oct;31(10):2287-94. doi: 10.1161/01.str.31.10.2287. PMID 11022052
- [Background] Kurl S, Tuomainen TP, Laukkanen JA, Nyyssonen K, Lakka T, Sivenius J, Salonen JT. Plasma vitamin C modifies the association between hypertension and risk of stroke. Stroke. 2002 Jun;33(6):1568-73. doi: 10.1161/01.str.0000017220.78722.d7. PMID 12052992
- [Background] Jacques PF, Sulsky SI, Perrone GE, Jenner J, Schaefer EJ. Effect of vitamin C supplementation on lipoprotein cholesterol, apolipoprotein, and triglyceride concentrations. Ann Epidemiol. 1995 Jan;5(1):52-9. doi: 10.1016/1047-2797(94)00041-q. PMID 7728285
- [Background] Simon JA, Hudes ES. Relation of serum ascorbic acid to serum lipids and lipoproteins in US adults. J Am Coll Nutr. 1998 Jun;17(3):250-5. doi: 10.1080/07315724.1998.10718755. PMID 9627911
- [Background] Moran JP, Cohen L, Greene JM, Xu G, Feldman EB, Hames CG, Feldman DS. Plasma ascorbic acid concentrations relate inversely to blood pressure in human subjects. Am J Clin Nutr. 1993 Feb;57(2):213-7. doi: 10.1093/ajcn/57.2.213. PMID 8424391
- [Background] McCarron DA, Morris CD, Henry HJ, Stanton JL. Blood pressure and nutrient intake in the United States. Science. 1984 Jun 29;224(4656):1392-8. doi: 10.1126/science.6729459.
- [Background] Carr AC, Shaw GM, Fowler AA, Natarajan R. Ascorbate-dependent vasopressor synthesis: a rationale for vitamin C administration in severe sepsis and septic shock? Crit Care. 2015 Nov 27;19:418. doi: 10.1186/s13054-015-1131-2. PMID 26612352
- [Background] Steinberg D, Parthasarathy S, Carew TE, Khoo JC, Witztum JL. Beyond cholesterol. Modifications of low-density lipoprotein that increase its atherogenicity. N Engl J Med. 1989 Apr 6;320(14):915-24. doi: 10.1056/NEJM198904063201407. No abstract available. PMID 2648148
- [Background] Armour J, Tyml K, Lidington D, Wilson JX. Ascorbate prevents microvascular dysfunction in the skeletal muscle of the septic rat. J Appl Physiol (1985). 2001 Mar;90(3):795-803. doi: 10.1152/jappl.2001.90.3.795. PMID 11181585
- [Background] Vahedi P, Rajabzadeh A, Soleimani A. An evaluation of the effects of ascorbic acid on the endothelium of coronary and aorta arteries in lead-intoxicated rabbits. SAGE Open Med. 2022 Jun 24;10:20503121221105330. doi: 10.1177/20503121221105330. eCollection 2022. PMID 35769490
- [Background] Solzbach U, Hornig B, Jeserich M, Just H. Vitamin C improves endothelial dysfunction of epicardial coronary arteries in hypertensive patients. Circulation. 1997 Sep 2;96(5):1513-9. doi: 10.1161/01.cir.96.5.1513. PMID 9315540
- [Background] Madokoro Y, Kamikokuryo C, Niiyama S, Ito T, Hara S, Ichinose H, Kakihana Y. Early ascorbic acid administration prevents vascular endothelial cell damage in septic mice. Front Pharmacol. 2022 Oct 6;13:929448. doi: 10.3389/fphar.2022.929448. eCollection 2022. PMID 36278212
- [Background] Vogiatzi G, Tousoulis D, Stefanadis C. The role of oxidative stress in atherosclerosis. Hellenic J Cardiol. 2009 Sep-Oct;50(5):402-9. No abstract available. PMID 19767282
- [Background] Batty M, Bennett MR, Yu E. The Role of Oxidative Stress in Atherosclerosis. Cells. 2022 Nov 30;11(23):3843. doi: 10.3390/cells11233843. PMID 36497101
- [Background] Chen Y, Luo X, Xu B, Bao X, Jia H, Yu B. Oxidative Stress-Mediated Programmed Cell Death: a Potential Therapy Target for Atherosclerosis. Cardiovasc Drugs Ther. 2024 Aug;38(4):819-832. doi: 10.1007/s10557-022-07414-z. Epub 2022 Dec 16. PMID 36522550
- [Background] Pacher P, Nivorozhkin A, Szabo C. Therapeutic effects of xanthine oxidase inhibitors: renaissance half a century after the discovery of allopurinol. Pharmacol Rev. 2006 Mar;58(1):87-114. doi: 10.1124/pr.58.1.6. PMID 16507884
- [Background] Connor M. Allopurinol for pain relief: more than just crystal clearance? Br J Pharmacol. 2009 Jan;156(1):4-6. doi: 10.1111/j.1476-5381.2008.00065.x. PMID 19133987
- [Background] Cavarocchi NC, England MD, O'Brien JF, Solis E, Russo P, Schaff HV, Orszulak TA, Pluth JR, Kaye MP. Superoxide generation during cardiopulmonary bypass: is there a role for vitamin E? J Surg Res. 1986 Jun;40(6):519-27. doi: 10.1016/0022-4804(86)90093-4. PMID 3018363
- [Background] Lassnigg A, Punz A, Barker R, Keznickl P, Manhart N, Roth E, Hiesmayr M. Influence of intravenous vitamin E supplementation in cardiac surgery on oxidative stress: a double-blinded, randomized, controlled study. Br J Anaesth. 2003 Feb;90(2):148-54. doi: 10.1093/bja/aeg042. PMID 12538369
- [Background] Valle-Giner I, Marti-Bonmati E, Alegria-Toran A, Montero A, Morcillo EJ. Changes in alpha-tocopherol and retinol levels during cardiopulmonary bypass correlate with maximal arterial partial pressure of oxygen. Free Radic Res. 2007 Sep;41(9):1061-7. doi: 10.1080/10715760701466389. PMID 17729125
- [Background] Westhuyzen J, Cochrane AD, Tesar PJ, Mau T, Cross DB, Frenneaux MP, Khafagi FA, Fleming SJ. Effect of preoperative supplementation with alpha-tocopherol and ascorbic acid on myocardial injury in patients undergoing cardiac operations. J Thorac Cardiovasc Surg. 1997 May;113(5):942-8. doi: 10.1016/s0022-5223(97)70268-x. PMID 9159629
- [Background] Sisto T, Paajanen H, Metsa-Ketela T, Harmoinen A, Nordback I, Tarkka M. Pretreatment with antioxidants and allopurinol diminishes cardiac onset events in coronary artery bypass grafting. Ann Thorac Surg. 1995 Jun;59(6):1519-23. doi: 10.1016/0003-4975(95)00197-s. PMID 7771834
- [Background] Samadikhah J, Golzari SE, Sabermarouf B, Karimzadeh I, Tizro P, Mohammad Khanli H, Ghabili K. Efficacy of Combination Therapy of Statin and Vitamin C in Comparison with Statin in the Prevention of Post-CABG Atrial Fibrillation. Adv Pharm Bull. 2014;4(1):97-100. doi: 10.5681/apb.2014.015. Epub 2013 Dec 23. PMID 24409416
- [Background] Safaei N, Babaei H, Azarfarin R, Jodati AR, Yaghoubi A, Sheikhalizadeh MA. Comparative effect of grape seed extract (Vitis vinifera) and ascorbic acid in oxidative stress induced by on-pump coronary artery bypass surgery. Ann Card Anaesth. 2017 Jan-Mar;20(1):45-51. doi: 10.4103/0971-9784.197834. PMID 28074795
- [Background] Papoulidis P, Ananiadou O, Chalvatzoulis E, Ampatzidou F, Koutsogiannidis C, Karaiskos T, Madesis A, Drossos G. The role of ascorbic acid in the prevention of atrial fibrillation after elective on-pump myocardial revascularization surgery: a single-center experience--a pilot study. Interact Cardiovasc Thorac Surg. 2011 Feb;12(2):121-4. doi: 10.1510/icvts.2010.240473. Epub 2010 Nov 23. PMID 21098510
- [Background] Knodell RG, Tate MA, Akl BF, Wilson JW. Vitamin C prophylaxis for posttransfusion hepatitis: lack of effect in a controlled trial. Am J Clin Nutr. 1981 Jan;34(1):20-3. doi: 10.1093/ajcn/34.1.20. PMID 7446455
- [Background] Jouybar R, Kabgani H, Kamalipour H, et al. The perioperative effect of ascorbic acid on inflammatory response in coronary artery bypass graft surgery; a randomized controlled trial coronary artery bypass graft surgery. Iran Cardiovasc Res J 2012;6:13-17.
- [Background] Gunes T, Bozok S, Kestelli M, Yurekli I, Ilhan G, Ozpak B, Bademci M, Ozcem B, Sahin A. alpha-tocopherol and ascorbic acid in early postoperative period of cardiopulmonary bypass. J Cardiovasc Med (Hagerstown). 2012 Nov;13(11):691-9. doi: 10.2459/JCM.0b013e328356a2dc. PMID 22885531
- [Background] Eslami M, Badkoubeh RS, Mousavi M, Radmehr H, Salehi M, Tavakoli N, Avadi MR. Oral ascorbic acid in combination with beta-blockers is more effective than beta-blockers alone in the prevention of atrial fibrillation after coronary artery bypass grafting. Tex Heart Inst J. 2007;34(3):268-74. PMID 17948074
- [Background] Dehghani MR, Majidi N, Rahmani A, Asgari B, Rezaei Y. Effect of oral vitamin C on atrial fibrillation development after isolated coronary artery bypass grafting surgery: A prospective randomized clinical trial. Cardiol J. 2014;21(5):492-9. doi: 10.5603/CJ.a2013.0154. Epub 2013 Dec 2. PMID 24293167
- [Background] Das D, Sen C, Goswami A. Effect of Vitamin C on adrenal suppression by etomidate induction in patients undergoing cardiac surgery: A randomized controlled trial. Ann Card Anaesth. 2016 Jul-Sep;19(3):410-7. doi: 10.4103/0971-9784.185522. PMID 27397444
- [Background] Colby JA, Chen WT, Baker WL, Coleman CI, Reinhart K, Kluger J, White CM. Effect of ascorbic acid on inflammatory markers after cardiothoracic surgery. Am J Health Syst Pharm. 2011 Sep 1;68(17):1632-9. doi: 10.2146/ajhp100703. PMID 21856809
- [Background] Carnes CA, Chung MK, Nakayama T, Nakayama H, Baliga RS, Piao S, Kanderian A, Pavia S, Hamlin RL, McCarthy PM, Bauer JA, Van Wagoner DR. Ascorbate attenuates atrial pacing-induced peroxynitrite formation and electrical remodeling and decreases the incidence of postoperative atrial fibrillation. Circ Res. 2001 Sep 14;89(6):E32-8. doi: 10.1161/hh1801.097644. PMID 11557745
- [Background] Bjordahl PM, Helmer SD, Gosnell DJ, Wemmer GE, O'Hara WW, Milfeld DJ. Perioperative supplementation with ascorbic acid does not prevent atrial fibrillation in coronary artery bypass graft patients. Am J Surg. 2012 Dec;204(6):862-7; discussion 867. doi: 10.1016/j.amjsurg.2012.03.012. Epub 2012 Sep 28. PMID 23022248
- [Background] Antonic M. Effect of Ascorbic Acid on Postoperative Acute Kidney Injury in Coronary Artery Bypass Graft Patients: A Pilot Study. Heart Surg Forum. 2017 Oct 24;20(5):E214-E218. doi: 10.1532/hsf.1811. PMID 29087285
- [Background] Antonic M, Lipovec R, Gregorcic F, Juric P, Kosir G. Perioperative ascorbic acid supplementation does not reduce the incidence of postoperative atrial fibrillation in on-pump coronary artery bypass graft patients. J Cardiol. 2017 Jan;69(1):98-102. doi: 10.1016/j.jjcc.2016.01.010. Epub 2016 Feb 23. PMID 26917198
- [Background] Angdin M, Settergren G, Starkopf J, Zilmer M, Zilmer K, Vaage J. Protective effect of antioxidants on pulmonary endothelial function after cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 2003 Jun;17(3):314-20. doi: 10.1016/s1053-0770(03)00053-3. PMID 12827578
- [Background] Hill A, Clasen KC, Wendt S, Majoros AG, Stoppe C, Adhikari NKJ, Heyland DK, Benstoem C. Effects of Vitamin C on Organ Function in Cardiac Surgery Patients: A Systematic Review and Meta-Analysis. Nutrients. 2019 Sep 4;11(9):2103. doi: 10.3390/nu11092103. PMID 31487905
- [Background] Oktar GL, Sinci V, Kalaycioglu S, Soncul H, Gokgoz L, Halit V, Ersoz A. Biochemical and hemodynamic effects of ascorbic acid and alpha-tocopherol in coronary artery surgery. Scand J Clin Lab Invest. 2001;61(8):621-9. doi: 10.1080/003655101753267982. PMID 11768322
- [Background] Ballmer PE, Reinhart WH, Jordan P, Buhler E, Moser UK, Gey KF. Depletion of plasma vitamin C but not of vitamin E in response to cardiac operations. J Thorac Cardiovasc Surg. 1994 Aug;108(2):311-20. PMID 8041179
- [Background] Tai YH, Wu HL, Chu YH, Huang CH, Ho ST, Lin TC, Lu CC. Vitamin C supplementation attenuates oxidative stress and improves erythrocyte deformability in cardiac surgery with cardiopulmonary bypass. Chin J Physiol. 2022 Sep-Oct;65(5):241-249. doi: 10.4103/0304-4920.358234. PMID 36308079
- [Background] Rodemeister S, Duquesne M, Adolph M, Nohr D, Biesalski HK, Unertl K. Massive and long-lasting decrease in vitamin C plasma levels as a consequence of extracorporeal circulation. Nutrition. 2014 Jun;30(6):673-8. doi: 10.1016/j.nut.2013.10.026. Epub 2013 Nov 6. PMID 24631388
- [Background] Carr AC, Vissers MC, Cook JS. The effect of intravenous vitamin C on cancer- and chemotherapy-related fatigue and quality of life. Front Oncol. 2014 Oct 16;4:283. doi: 10.3389/fonc.2014.00283. eCollection 2014. PMID 25360419
- [Background] German Nutrition Society (DGE). New Reference Values for Vitamin C Intake. Ann Nutr Metab. 2015;67(1):13-20. doi: 10.1159/000434757. Epub 2015 Jul 22. PMID 26227083
- [Background] Hill A, Borgs C, Fitzner C, Stoppe C. Perioperative Vitamin C and E levels in Cardiac Surgery Patients and Their Clinical Significance. Nutrients. 2019 Sep 9;11(9):2157. doi: 10.3390/nu11092157. PMID 31505814
- [Background] Fukushima R, Yamazaki E. Vitamin C requirement in surgical patients. Curr Opin Clin Nutr Metab Care. 2010 Nov;13(6):669-76. doi: 10.1097/MCO.0b013e32833e05bc. PMID 20689415
- [Background] Rowe S, Carr AC. Global Vitamin C Status and Prevalence of Deficiency: A Cause for Concern? Nutrients. 2020 Jul 6;12(7):2008. doi: 10.3390/nu12072008. PMID 32640674
- [Background] Evans RM, Currie L, Campbell A. The distribution of ascorbic acid between various cellular components of blood, in normal individuals, and its relation to the plasma concentration. Br J Nutr. 1982 May;47(3):473-82. doi: 10.1079/bjn19820059. PMID 7082619
- [Background] Rumelin A, Jaehde U, Kerz T, Roth W, Kramer M, Fauth U. Early postoperative substitution procedure of the antioxidant ascorbic acid. J Nutr Biochem. 2005 Feb;16(2):104-8. doi: 10.1016/j.jnutbio.2004.10.005. PMID 15681169
- [Background] Carr AC, Rosengrave PC, Bayer S, Chambers S, Mehrtens J, Shaw GM. Hypovitaminosis C and vitamin C deficiency in critically ill patients despite recommended enteral and parenteral intakes. Crit Care. 2017 Dec 11;21(1):300. doi: 10.1186/s13054-017-1891-y. PMID 29228951
- [Background] Ellinger S, Stehle P. Efficacy of vitamin supplementation in situations with wound healing disorders: results from clinical intervention studies. Curr Opin Clin Nutr Metab Care. 2009 Nov;12(6):588-95. doi: 10.1097/MCO.0b013e328331a5b5. PMID 19770648
- [Background] Beattie AD, Sherlock S. Ascorbic acid deficiency in liver disease. Gut. 1976 Aug;17(8):571-5. doi: 10.1136/gut.17.8.571. PMID 976794
- [Background] Ginter E. Chronic marginal vitamin C deficiency: biochemistry and pathophysiology. World Rev Nutr Diet. 1979;33:104-41. doi: 10.1159/000402551. No abstract available. PMID 392953
- [Background] Ghalibaf MHE, Kianian F, Beigoli S, Behrouz S, Marefati N, Boskabady M, Boskabady MH. The effects of vitamin C on respiratory, allergic and immunological diseases: an experimental and clinical-based review. Inflammopharmacology. 2023 Apr;31(2):653-672. doi: 10.1007/s10787-023-01169-1. Epub 2023 Feb 27. PMID 36849854
- [Background] Otocka-Kmiecik A, Krol A. The Role of Vitamin C in Two Distinct Physiological States: Physical Activity and Sleep. Nutrients. 2020 Dec 21;12(12):3908. doi: 10.3390/nu12123908. PMID 33371359
- [Background] Tveden-Nyborg P. Vitamin C Deficiency in the Young Brain-Findings from Experimental Animal Models. Nutrients. 2021 May 15;13(5):1685. doi: 10.3390/nu13051685. PMID 34063417
- [Background] Nowak D. Vitamin C in Human Health and Disease. Nutrients. 2021 May 11;13(5):1595. doi: 10.3390/nu13051595. PMID 34064549
- [Background] Dosedel M, Jirkovsky E, Macakova K, Krcmova LK, Javorska L, Pourova J, Mercolini L, Remiao F, Novakova L, Mladenka P, On Behalf Of The Oemonom. Vitamin C-Sources, Physiological Role, Kinetics, Deficiency, Use, Toxicity, and Determination. Nutrients. 2021 Feb 13;13(2):615. doi: 10.3390/nu13020615. PMID 33668681
- [Background] Nyyssonen K, Parviainen MT, Salonen R, Tuomilehto J, Salonen JT. Vitamin C deficiency and risk of myocardial infarction: prospective population study of men from eastern Finland. BMJ. 1997 Mar 1;314(7081):634-8. doi: 10.1136/bmj.314.7081.634. PMID 9066474
- [Background] Kristenson M, Zieden B, Kucinskiene Z, Elinder LS, Bergdahl B, Elwing B, Abaravicius A, Razinkoviene L, Calkauskas H, Olsson AG. Antioxidant state and mortality from coronary heart disease in Lithuanian and Swedish men: concomitant cross sectional study of men aged 50. BMJ. 1997 Mar 1;314(7081):629-33. doi: 10.1136/bmj.314.7081.629. PMID 9066473
- [Background] Al-Khudairy L, Flowers N, Wheelhouse R, Ghannam O, Hartley L, Stranges S, Rees K. Vitamin C supplementation for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2017 Mar 16;3(3):CD011114. doi: 10.1002/14651858.CD011114.pub2. PMID 28301692
- [Background] National Center for Biotechnology Information . PubChem Compound Summary for CID 54670067, Ascorbic Acid. Accessed Oct. 29 https://pubchem.ncbi.nlm.nih.gov/compound/Ascorbic-Acid, 2023.
- [Background] Morelli MB, Gambardella J, Castellanos V, Trimarco V, Santulli G. Vitamin C and Cardiovascular Disease: An Update. Antioxidants (Basel). 2020 Dec 3;9(12):1227. doi: 10.3390/antiox9121227. PMID 33287462
- [Background] Naidu KA. Vitamin C in human health and disease is still a mystery? An overview. Nutr J. 2003 Aug 21;2:7. doi: 10.1186/1475-2891-2-7. PMID 14498993
- [Background] Mandl J, Szarka A, Banhegyi G. Vitamin C: update on physiology and pharmacology. Br J Pharmacol. 2009 Aug;157(7):1097-110. doi: 10.1111/j.1476-5381.2009.00282.x. Epub 2009 Jun 5. PMID 19508394
- [Background] Paciolla C, Fortunato S, Dipierro N, Paradiso A, De Leonardis S, Mastropasqua L, de Pinto MC. Vitamin C in Plants: From Functions to Biofortification. Antioxidants (Basel). 2019 Oct 29;8(11):519. doi: 10.3390/antiox8110519. PMID 31671820
- [Background] Njus D, Kelley PM, Tu YJ, Schlegel HB. Ascorbic acid: The chemistry underlying its antioxidant properties. Free Radic Biol Med. 2020 Nov 1;159:37-43. doi: 10.1016/j.freeradbiomed.2020.07.013. Epub 2020 Jul 30. PMID 32738399
- [Background] May MJ, Vernoux T, Leaver C, et al. Glutathione homeostasis in plants: implications for environmental sensing and plant development. J Exp Bot 1998;49:649-667.
- [Background] Zechmann B. Compartment-specific importance of glutathione during abiotic and biotic stress. Front Plant Sci. 2014 Oct 20;5:566. doi: 10.3389/fpls.2014.00566. eCollection 2014. PMID 25368627
- [Background] May JM, Harrison FE. Role of vitamin C in the function of the vascular endothelium. Antioxid Redox Signal. 2013 Dec 10;19(17):2068-83. doi: 10.1089/ars.2013.5205. Epub 2013 May 29. PMID 23581713
- [Background] Dingchao H, Zhiduan Q, Liye H, Xiaodong F. The protective effects of high-dose ascorbic acid on myocardium against reperfusion injury during and after cardiopulmonary bypass. Thorac Cardiovasc Surg. 1994 Oct;42(5):276-8. doi: 10.1055/s-2007-1016504. PMID 7863489
- [Background] Winkler BS, Orselli SM, Rex TS. The redox couple between glutathione and ascorbic acid: a chemical and physiological perspective. Free Radic Biol Med. 1994 Oct;17(4):333-49. doi: 10.1016/0891-5849(94)90019-1. PMID 8001837
- [Background] Rodrigo R, Guichard C, Charles R. Clinical pharmacology and therapeutic use of antioxidant vitamins. Fundam Clin Pharmacol. 2007 Apr;21(2):111-27. doi: 10.1111/j.1472-8206.2006.00466.x. PMID 17391284
- [Background] Yussif NM. Vitamin C - an update on current uses and functions. Vitam C - an Updat Curr Uses Funct 2019;1:7-8.
- [Background] Sadeghpour A, Alizadehasl A, Kyavar M, Sadeghi T, Moludi J, Gholizadeh F, Totonchi Z, Ghadrdoost B. Impact of vitamin C supplementation on post-cardiac surgery ICU and hospital length of stay. Anesth Pain Med. 2015 Feb 19;5(1):e25337. doi: 10.5812/aapm.25337. eCollection 2015 Feb. PMID 25789244
- [Background] Fernandes GS, Fernandez CD, Campos KE, Damasceno DC, Anselmo-Franci JA, Kempinas WD. Vitamin C partially attenuates male reproductive deficits in hyperglycemic rats. Reprod Biol Endocrinol. 2011 Jul 27;9:100. doi: 10.1186/1477-7827-9-100. PMID 21794102
- [Background] Sonmez M, Turk G, Yuce A. The effect of ascorbic acid supplementation on sperm quality, lipid peroxidation and testosterone levels of male Wistar rats. Theriogenology. 2005 Apr 15;63(7):2063-72. doi: 10.1016/j.theriogenology.2004.10.003. Epub 2004 Nov 18. PMID 15823361
- [Background] Holford P, Carr AC, Jovic TH, Ali SR, Whitaker IS, Marik PE, Smith AD. Vitamin C-An Adjunctive Therapy for Respiratory Infection, Sepsis and COVID-19. Nutrients. 2020 Dec 7;12(12):3760. doi: 10.3390/nu12123760. PMID 33297491
- [Background] Paltiel O, Gordon L, Berg D, Israeli A. Effect of a computerized alert on the management of hypokalemia in hospitalized patients. Arch Intern Med. 2003 Jan 27;163(2):200-4. doi: 10.1001/archinte.163.2.200. PMID 12546610
- [Background] Geng J, Qian J, Si W, Cheng H, Ji F, Shen Z. The clinical benefits of perioperative antioxidant vitamin therapy in patients undergoing cardiac surgery: a meta-analysis. Interact Cardiovasc Thorac Surg. 2017 Dec 1;25(6):966-974. doi: 10.1093/icvts/ivx178. PMID 28645181
- [Background] Zhu YB, Zhang YP, Zhang J, Zhang YB. Evaluation of Vitamin C Supplementation on Kidney Function and Vascular Reactivity Following Renal Ischemic Injury in Mice. Kidney Blood Press Res. 2016;41(4):460-70. doi: 10.1159/000443447. Epub 2016 Jul 15. PMID 27415798
- [Background] Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. Arch Surg. 2000 Mar;135(3):326-31. doi: 10.1001/archsurg.135.3.326. PMID 10722036
- [Background] Kahn SA, Beers RJ, Lentz CW. Resuscitation after severe burn injury using high-dose ascorbic acid: a retrospective review. J Burn Care Res. 2011 Jan-Feb;32(1):110-7. doi: 10.1097/BCR.0b013e318204b336. PMID 21131846
- [Background] Travica N, Ried K, Sali A, Scholey A, Hudson I, Pipingas A. Vitamin C Status and Cognitive Function: A Systematic Review. Nutrients. 2017 Aug 30;9(9):960. doi: 10.3390/nu9090960. PMID 28867798
- [Background] Eldridge CF, Bunge MB, Bunge RP, Wood PM. Differentiation of axon-related Schwann cells in vitro. I. Ascorbic acid regulates basal lamina assembly and myelin formation. J Cell Biol. 1987 Aug;105(2):1023-34. doi: 10.1083/jcb.105.2.1023. PMID 3624305
- [Background] Huang J, Agus DB, Winfree CJ, Kiss S, Mack WJ, McTaggart RA, Choudhri TF, Kim LJ, Mocco J, Pinsky DJ, Fox WD, Israel RJ, Boyd TA, Golde DW, Connolly ES Jr. Dehydroascorbic acid, a blood-brain barrier transportable form of vitamin C, mediates potent cerebroprotection in experimental stroke. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):11720-4. doi: 10.1073/pnas.171325998. PMID 11573006
- [Background] Berger MM, Oudemans-van Straaten HM. Vitamin C supplementation in the critically ill patient. Curr Opin Clin Nutr Metab Care. 2015 Mar;18(2):193-201. doi: 10.1097/MCO.0000000000000148. PMID 25635594
- [Background] Oakes B, Bolia IK, Weber AE, Petrigliano FA. Vitamin C in orthopedic practices: Current concepts, novel ideas, and future perspectives. J Orthop Res. 2021 Apr;39(4):698-706. doi: 10.1002/jor.24947. Epub 2021 Jan 4. PMID 33300201
- [Background] Brzezinska O, Lukasik Z, Makowska J, Walczak K. Role of Vitamin C in Osteoporosis Development and Treatment-A Literature Review. Nutrients. 2020 Aug 10;12(8):2394. doi: 10.3390/nu12082394. PMID 32785080
- [Background] Levine M, Rumsey SC, Daruwala R, Park JB, Wang Y. Criteria and recommendations for vitamin C intake. JAMA. 1999 Apr 21;281(15):1415-23. doi: 10.1001/jama.281.15.1415. PMID 10217058
- [Background] Yamamoto T, Kinoshita M, Shinomiya N, Hiroi S, Sugasawa H, Matsushita Y, Majima T, Saitoh D, Seki S. Pretreatment with ascorbic acid prevents lethal gastrointestinal syndrome in mice receiving a massive amount of radiation. J Radiat Res. 2010;51(2):145-56. doi: 10.1269/jrr.09078. Epub 2009 Dec 4. PMID 19959877
- [Background] Al-Asmari AK, Khan AQ, Al-Qasim AM, Al-Yousef Y. Ascorbic acid attenuates antineoplastic drug 5-fluorouracil induced gastrointestinal toxicity in rats by modulating the expression of inflammatory mediators. Toxicol Rep. 2015 Jun 15;2:908-916. doi: 10.1016/j.toxrep.2015.06.006. eCollection 2015. PMID 28962429
- [Background] Pullar JM, Carr AC, Vissers MCM. The Roles of Vitamin C in Skin Health. Nutrients. 2017 Aug 12;9(8):866. doi: 10.3390/nu9080866. PMID 28805671
- [Background] Carr AC, Maggini S. Vitamin C and Immune Function. Nutrients. 2017 Nov 3;9(11):1211. doi: 10.3390/nu9111211. PMID 29099763
- [Background] Lim JC, Caballero Arredondo M, Braakhuis AJ, Donaldson PJ. Vitamin C and the Lens: New Insights into Delaying the Onset of Cataract. Nutrients. 2020 Oct 14;12(10):3142. doi: 10.3390/nu12103142. PMID 33066702
- [Background] Grosso G, Bei R, Mistretta A, Marventano S, Calabrese G, Masuelli L, Giganti MG, Modesti A, Galvano F, Gazzolo D. Effects of vitamin C on health: a review of evidence. Front Biosci (Landmark Ed). 2013 Jun 1;18(3):1017-29. doi: 10.2741/4160. PMID 23747864
- [Background] Moser MA, Chun OK. Vitamin C and Heart Health: A Review Based on Findings from Epidemiologic Studies. Int J Mol Sci. 2016 Aug 12;17(8):1328. doi: 10.3390/ijms17081328. PMID 27529239
- [Background] Chambial S, Dwivedi S, Shukla KK, John PJ, Sharma P. Vitamin C in disease prevention and cure: an overview. Indian J Clin Biochem. 2013 Oct;28(4):314-28. doi: 10.1007/s12291-013-0375-3. Epub 2013 Sep 1. PMID 24426232
- [Background] Juraschek SP, Guallar E, Appel LJ, Miller ER 3rd. Effects of vitamin C supplementation on blood pressure: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2012 May;95(5):1079-88. doi: 10.3945/ajcn.111.027995. Epub 2012 Apr 4. PMID 22492364
- [Background] Hill A, Wendt S, Benstoem C, Neubauer C, Meybohm P, Langlois P, Adhikari NK, Heyland DK, Stoppe C. Vitamin C to Improve Organ Dysfunction in Cardiac Surgery Patients-Review and Pragmatic Approach. Nutrients. 2018 Jul 27;10(8):974. doi: 10.3390/nu10080974. PMID 30060468
- [Background] Wilson JX. Evaluation of vitamin C for adjuvant sepsis therapy. Antioxid Redox Signal. 2013 Dec 10;19(17):2129-40. doi: 10.1089/ars.2013.5401. Epub 2013 Jun 25. PMID 23682970
- [Background] Tyml K. Vitamin C and Microvascular Dysfunction in Systemic Inflammation. Antioxidants (Basel). 2017 Jun 29;6(3):49. doi: 10.3390/antiox6030049. PMID 28661424
- [Background] Takahashi T, Lord B, Schulze PC, Fryer RM, Sarang SS, Gullans SR, Lee RT. Ascorbic acid enhances differentiation of embryonic stem cells into cardiac myocytes. Circulation. 2003 Apr 15;107(14):1912-6. doi: 10.1161/01.CIR.0000064899.53876.A3. Epub 2003 Mar 31. PMID 12668514
- [Background] Ashor AW, Siervo M, Lara J, Oggioni C, Mathers JC. Antioxidant vitamin supplementation reduces arterial stiffness in adults: a systematic review and meta-analysis of randomized controlled trials. J Nutr. 2014 Oct;144(10):1594-602. doi: 10.3945/jn.114.195826. Epub 2014 Aug 6. PMID 25098780
- [Background] Ashor AW, Lara J, Mathers JC, Siervo M. Effect of vitamin C on endothelial function in health and disease: a systematic review and meta-analysis of randomised controlled trials. Atherosclerosis. 2014 Jul;235(1):9-20. doi: 10.1016/j.atherosclerosis.2014.04.004. Epub 2014 Apr 18. PMID 24792921
- [Background] Hu X, Yuan L, Wang H, Li C, Cai J, Hu Y, Ma C. Efficacy and safety of vitamin C for atrial fibrillation after cardiac surgery: A meta-analysis with trial sequential analysis of randomized controlled trials. Int J Surg. 2017 Jan;37:58-64. doi: 10.1016/j.ijsu.2016.12.009. Epub 2016 Dec 9. PMID 27956113
- [Background] Polymeropoulos E, Bagos P, Papadimitriou M, Rizos I, Patsouris E, Tauoumpoulis I. Vitamin C for the Prevention of Postoperative Atrial Fibrillation after Cardiac Surgery: A Meta-Analysis. Adv Pharm Bull. 2016 Jun;6(2):243-50. doi: 10.15171/apb.2016.033. Epub 2016 Jun 30. PMID 27478787
- [Background] Tsao CS. An overview of ascorbic acid chemistry and biochemistry. In: Packer L, Fuchs JE, eds. Vitamin C in Health and Disease. Marcel Dekker Inc; 1997:25-58.
- [Background] Zabet MH, Mohammadi M, Ramezani M, Khalili H. Effect of high-dose Ascorbic acid on vasopressor's requirement in septic shock. J Res Pharm Pract. 2016 Apr-Jun;5(2):94-100. doi: 10.4103/2279-042X.179569. PMID 27162802
- [Background] Spoelstra-de Man AME, Elbers PWG, Oudemans-van Straaten HM. Making sense of early high-dose intravenous vitamin C in ischemia/reperfusion injury. Crit Care. 2018 Mar 20;22(1):70. doi: 10.1186/s13054-018-1996-y. PMID 29558975
- [Background] Oudemans-van Straaten HM, Spoelstra-de Man AM, de Waard MC. Vitamin C revisited. Crit Care. 2014 Aug 6;18(4):460. doi: 10.1186/s13054-014-0460-x. PMID 25185110
- [Background] Odgaard-Jensen J, Vist GE, Timmer A, Kunz R, Akl EA, Schunemann H, Briel M, Nordmann AJ, Pregno S, Oxman AD. Randomisation to protect against selection bias in healthcare trials. Cochrane Database Syst Rev. 2011 Apr 13;2011(4):MR000012. doi: 10.1002/14651858.MR000012.pub3. PMID 21491415
- [Background] Schulz KF, Chalmers I, Hayes RJ, Altman DG. Empirical evidence of bias. Dimensions of methodological quality associated with estimates of treatment effects in controlled trials. JAMA. 1995 Feb 1;273(5):408-12. doi: 10.1001/jama.273.5.408. PMID 7823387
- [Background] Day SJ, Altman DG. Statistics notes: blinding in clinical trials and other studies. BMJ. 2000 Aug 19-26;321(7259):504. doi: 10.1136/bmj.321.7259.504. No abstract available. PMID 10948038
- [Background] Kane SP. Sample Size Calculator. ClinCalc: https://clincalc.com/stats/samplesize.aspx. Updated July 24, 2019. Accessed August 4, 2021.
- [Background] Rosner, Bernard (Bernard A.). (2011). Fundamentals of biostatistics. Boston :Brooks/Cole, Cengage Learning.
- [Background] Hulley SB, Cummings SR, Browner WS, Grady D, Newman TB. Designing clinical research : an epidemiologic approach. 4th ed. Philadelphia, PA: Lippincott Williams & Wilkins; 2013. Appendix 6A, page 73. ISBN/ISSN: 9781608318049
- [Background] Nielsen SJ, Karlsson M, Bjorklund E, Martinsson A, Hansson EC, Malm CJ, Pivodic A, Jeppsson A. Socioeconomic Factors, Secondary Prevention Medication, and Long-Term Survival After Coronary Artery Bypass Grafting: A Population-Based Cohort Study From the SWEDEHEART Registry. J Am Heart Assoc. 2020 Mar 3;9(5):e015491. doi: 10.1161/JAHA.119.015491. Epub 2020 Mar 2. PMID 32114890
- [Background] Farkouh ME, Domanski M, Dangas GD, Godoy LC, Mack MJ, Siami FS, Hamza TH, Shah B, Stefanini GG, Sidhu MS, Tanguay JF, Ramanathan K, Sharma SK, French J, Hueb W, Cohen DJ, Fuster V; FREEDOM Follow-On Study Investigators. Long-Term Survival Following Multivessel Revascularization in Patients With Diabetes: The FREEDOM Follow-On Study. J Am Coll Cardiol. 2019 Feb 19;73(6):629-638. doi: 10.1016/j.jacc.2018.11.001. Epub 2018 Nov 11. PMID 30428398
- [Background] Head SJ, Milojevic M, Daemen J, Ahn JM, Boersma E, Christiansen EH, Domanski MJ, Farkouh ME, Flather M, Fuster V, Hlatky MA, Holm NR, Hueb WA, Kamalesh M, Kim YH, Makikallio T, Mohr FW, Papageorgiou G, Park SJ, Rodriguez AE, Sabik JF 3rd, Stables RH, Stone GW, Serruys PW, Kappetein AP. Mortality after coronary artery bypass grafting versus percutaneous coronary intervention with stenting for coronary artery disease: a pooled analysis of individual patient data. Lancet. 2018 Mar 10;391(10124):939-948. doi: 10.1016/S0140-6736(18)30423-9. Epub 2018 Feb 23. PMID 29478841
- [Background] Xenogiannis I, Tajti P, Hall AB, Alaswad K, Rinfret S, Nicholson W, Karmpaliotis D, Mashayekhi K, Furkalo S, Cavalcante JL, Burke MN, Brilakis ES. Update on Cardiac Catheterization in Patients With Prior Coronary Artery Bypass Graft Surgery. JACC Cardiovasc Interv. 2019 Sep 9;12(17):1635-1649. doi: 10.1016/j.jcin.2019.04.051. Epub 2019 Aug 14. PMID 31422085
- [Background] Doenst T, Haverich A, Serruys P, Bonow RO, Kappetein P, Falk V, Velazquez E, Diegeler A, Sigusch H. PCI and CABG for Treating Stable Coronary Artery Disease: JACC Review Topic of the Week. J Am Coll Cardiol. 2019 Mar 5;73(8):964-976. doi: 10.1016/j.jacc.2018.11.053. PMID 30819365
- [Background] Bjorklund E, Nielsen SJ, Hansson EC, Karlsson M, Wallinder A, Martinsson A, Tygesen H, Romlin BS, Malm CJ, Pivodic A, Jeppsson A. Secondary prevention medications after coronary artery bypass grafting and long-term survival: a population-based longitudinal study from the SWEDEHEART registry. Eur Heart J. 2020 May 1;41(17):1653-1661. doi: 10.1093/eurheartj/ehz714. PMID 31638654
- [Background] Watson D, O'Connell Motherway M, Schoterman MH, van Neerven RJ, Nauta A, van Sinderen D. Selective carbohydrate utilization by lactobacilli and bifidobacteria. J Appl Microbiol. 2013 Apr;114(4):1132-46. doi: 10.1111/jam.12105. Epub 2013 Jan 11. PMID 23240984
- [Background] K. Tuohy, C. Ziemer, A. Klinder, Y. Knobel, B. Pool-Zobel and G. Gibson, "A Human Volunteer Study to Determine the Prebiotic Effects of Lactulose Powder on Human Colonic Microbiota.," Microbial Ecology in Health and Disease, vol. 14, no. 3, 2011.
- [Background] Markowiak P, Slizewska K. Effects of Probiotics, Prebiotics, and Synbiotics on Human Health. Nutrients. 2017 Sep 15;9(9):1021. doi: 10.3390/nu9091021. PMID 28914794
- [Background] Slavin J. Fiber and prebiotics: mechanisms and health benefits. Nutrients. 2013 Apr 22;5(4):1417-35. doi: 10.3390/nu5041417. PMID 23609775
- [Background] Roberfroid M. Prebiotics: the concept revisited. J Nutr. 2007 Mar;137(3 Suppl 2):830S-7S. doi: 10.1093/jn/137.3.830S. PMID 17311983
- [Background] Cardelle-Cobas A, Corzo N, Olano A, Pelaez C, Requena T, Avila M. Galactooligosaccharides derived from lactose and lactulose: influence of structure on Lactobacillus, Streptococcus and Bifidobacterium growth. Int J Food Microbiol. 2011 Sep 1;149(1):81-7. doi: 10.1016/j.ijfoodmicro.2011.05.026. Epub 2011 Jun 12. PMID 21700354
- [Background] Musa MA, Kabir M, Hossain MI, Ahmed E, Siddique A, Rashid H, Mahfuz M, Mondal D, Ahmed T, Petri WA, Haque R. Measurement of intestinal permeability using lactulose and mannitol with conventional five hours and shortened two hours urine collection by two different methods: HPAE-PAD and LC-MSMS. PLoS One. 2019 Aug 8;14(8):e0220397. doi: 10.1371/journal.pone.0220397. eCollection 2019. PMID 31393913
- [Background] Nath A, Molnar MA, Csighy A, Koszegi K, Galambos I, Huszar KP, Koris A, Vatai G. Biological Activities of Lactose-Based Prebiotics and Symbiosis with Probiotics on Controlling Osteoporosis, Blood-Lipid and Glucose Levels. Medicina (Kaunas). 2018 Dec 3;54(6):98. doi: 10.3390/medicina54060098. PMID 30513975
- [Background] Nath A, Haktanirlar G, Varga A, Molnar MA, Albert K, Galambos I, Koris A, Vatai G. Biological Activities of Lactose-Derived Prebiotics and Symbiotic with Probiotics on Gastrointestinal System. Medicina (Kaunas). 2018 Apr 17;54(2):18. doi: 10.3390/medicina54020018. PMID 30344249
- [Background] Zhai S, Zhu L, Qin S, Li L. Effect of lactulose intervention on gut microbiota and short chain fatty acid composition of C57BL/6J mice. Microbiologyopen. 2018 Dec;7(6):e00612. doi: 10.1002/mbo3.612. Epub 2018 Mar 24. PMID 29575825
- [Background] Bothe MK, Maathuis AJH, Bellmann S, van der Vossen JMBM, Berressem D, Koehler A, Schwejda-Guettes S, Gaigg B, Kuchinka-Koch A, Stover JF. Dose-Dependent Prebiotic Effect of Lactulose in a Computer-Controlled In Vitro Model of the Human Large Intestine. Nutrients. 2017 Jul 18;9(7):767. doi: 10.3390/nu9070767. PMID 28718839
- [Background] Ridola L, Faccioli J, Nardelli S, Gioia S, Riggio O. Hepatic Encephalopathy: Diagnosis and Management. J Transl Int Med. 2020 Dec 31;8(4):210-219. doi: 10.2478/jtim-2020-0034. eCollection 2020 Dec. PMID 33511048
- [Background] Pranami, D., Sharma, R., & Pathak, H. (2017). Lactulose: a prebiotic, laxative and detoxifying agent. Drugs & Therapy Perspectives, 33(5), 228-233.
- [Background] Fuller S, Beck E, Salman H, Tapsell L. New Horizons for the Study of Dietary Fiber and Health: A Review. Plant Foods Hum Nutr. 2016 Mar;71(1):1-12. doi: 10.1007/s11130-016-0529-6. PMID 26847187
- [Background] Žilić, S., Dodig, D., Milašinović-Šeremešić, M., Kandić, V., Kostadinović, M., Prodanović, S., & Savić, Đ. (2011). Small grain cereals compared for dietary fibre and protein contents. Genetika, 43(2), 381-395. https://doi.org/10.2298/GENSR1102381Z
- [Background] Mudgil D, Barak S. Composition, properties and health benefits of indigestible carbohydrate polymers as dietary fiber: a review. Int J Biol Macromol. 2013 Oct;61:1-6. doi: 10.1016/j.ijbiomac.2013.06.044. Epub 2013 Jul 2. PMID 23831534
- [Background] Modern enterosorbents and mechanisms of their action. Efferent therapy, 11(4), 3.
- [Background] A review on enterosorbents and their application in clinical practice: Removal of toxic metals Author links open overlay panelSevda Fatullayeva , Dilgam Tagiyev, Nizami Zeynalov
- [Background] Liu R, Dai L, Xu C, Wang K, Zheng C, Si C. Lignin-Based Micro- and Nanomaterials and their Composites in Biomedical Applications. ChemSusChem. 2020 Sep 7;13(17):4266-4283. doi: 10.1002/cssc.202000783. Epub 2020 Jun 25. PMID 32462781
- [Background] Ismailova, M. G., Yunuskhodjaeva, K. G., & Boyko, P. L. I. I. B. (2014). Physical-chemical and pharmacological research on new lignin enterosorbent. Journal of Pharmacy and Pharmacology, 2, 642-651.
- [Background] Kumar R, Butreddy A, Kommineni N, Reddy PG, Bunekar N, Sarkar C, Dutt S, Mishra VK, Aadil KR, Mishra YK, Oupicky D, Kaushik A. Lignin: Drug/Gene Delivery and Tissue Engineering Applications. Int J Nanomedicine. 2021 Mar 26;16:2419-2441. doi: 10.2147/IJN.S303462. eCollection 2021. PMID 33814908
- [Background] Saravanan P, Davidson NC, Schmidt EB, Calder PC. Cardiovascular effects of marine omega-3 fatty acids. Lancet. 2010 Aug 14;376(9740):540-50. doi: 10.1016/S0140-6736(10)60445-X. Epub 2010 Jul 15. PMID 20638121
- [Background] Schmidt EB, Arnesen H, Christensen JH, Rasmussen LH, Kristensen SD, De Caterina R. Marine n-3 polyunsaturated fatty acids and coronary heart disease: Part II. clinical trials and recommendations. Thromb Res. 2005;115(4):257-62. doi: 10.1016/j.thromres.2004.09.007. No abstract available. PMID 15668184
- [Background] Arnesen H. n-3 fatty acids and revascularization procedures. Lipids. 2001;36 Suppl:S103-6. doi: 10.1007/s11745-001-0690-z. PMID 11837981
- [Background] Vijayakumar M, Vasudevan DM, Sundaram KR, Krishnan S, Vaidyanathan K, Nandakumar S, Chandrasekhar R, Mathew N. A randomized study of coconut oil versus sunflower oil on cardiovascular risk factors in patients with stable coronary heart disease. Indian Heart J. 2016 Jul-Aug;68(4):498-506. doi: 10.1016/j.ihj.2015.10.384. Epub 2016 Jan 13. PMID 27543472
- [Background] Raitt MH, Connor WE, Morris C, Kron J, Halperin B, Chugh SS, McClelland J, Cook J, MacMurdy K, Swenson R, Connor SL, Gerhard G, Kraemer DF, Oseran D, Marchant C, Calhoun D, Shnider R, McAnulty J. Fish oil supplementation and risk of ventricular tachycardia and ventricular fibrillation in patients with implantable defibrillators: a randomized controlled trial. JAMA. 2005 Jun 15;293(23):2884-91. doi: 10.1001/jama.293.23.2884. PMID 15956633
- [Background] Nye ER, Ablett MB, Robertson MC, Ilsley CD, Sutherland WH. Effect of eicosapentaenoic acid on restenosis rate, clinical course and blood lipids in patients after percutaneous transluminal coronary angioplasty. Aust N Z J Med. 1990 Aug;20(4):549-52. doi: 10.1111/j.1445-5994.1990.tb01311.x. PMID 2222347
- [Background] Sacks FM, Stone PH, Gibson CM, Silverman DI, Rosner B, Pasternak RC. Controlled trial of fish oil for regression of human coronary atherosclerosis. HARP Research Group. J Am Coll Cardiol. 1995 Jun;25(7):1492-8. doi: 10.1016/0735-1097(95)00095-l. PMID 7759696
- [Background] Danthiir V, Burns NR, Nettelbeck T, Wilson C, Wittert G. The older people, omega-3, and cognitive health (EPOCH) trial design and methodology: a randomised, double-blind, controlled trial investigating the effect of long-chain omega-3 fatty acids on cognitive ageing and wellbeing in cognitively healthy older adults. Nutr J. 2011 Oct 20;10:117. doi: 10.1186/1475-2891-10-117. PMID 22011460
- [Background] Doi M, Nosaka K, Miyoshi T, Iwamoto M, Kajiya M, Okawa K, Nakayama R, Takagi W, Takeda K, Hirohata S, Ito H. Early eicosapentaenoic acid treatment after percutaneous coronary intervention reduces acute inflammatory responses and ventricular arrhythmias in patients with acute myocardial infarction: a randomized, controlled study. Int J Cardiol. 2014 Oct 20;176(3):577-82. doi: 10.1016/j.ijcard.2014.08.055. Epub 2014 Aug 19. PMID 25305703
- [Background] Abdelhamid AS, Martin N, Bridges C, Brainard JS, Wang X, Brown TJ, Hanson S, Jimoh OF, Ajabnoor SM, Deane KH, Song F, Hooper L. Polyunsaturated fatty acids for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2018 Nov 27;11(11):CD012345. doi: 10.1002/14651858.CD012345.pub3. PMID 30484282
- [Background] Studer M, Briel M, Leimenstoll B, Glass TR, Bucher HC. Effect of different antilipidemic agents and diets on mortality: a systematic review. Arch Intern Med. 2005 Apr 11;165(7):725-30. doi: 10.1001/archinte.165.7.725. PMID 15824290
- [Background] Bucher HC, Hengstler P, Schindler C, Meier G. N-3 polyunsaturated fatty acids in coronary heart disease: a meta-analysis of randomized controlled trials. Am J Med. 2002 Mar;112(4):298-304. doi: 10.1016/s0002-9343(01)01114-7. PMID 11893369
- [Background] Dietary supplementation with n-3 polyunsaturated fatty acids and vitamin E after myocardial infarction: results of the GISSI-Prevenzione trial. Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto miocardico. Lancet. 1999 Aug 7;354(9177):447-55. PMID 10465168
- [Background] Lavie CJ, Milani RV, Mehra MR, Ventura HO. Omega-3 polyunsaturated fatty acids and cardiovascular diseases. J Am Coll Cardiol. 2009 Aug 11;54(7):585-94. doi: 10.1016/j.jacc.2009.02.084. PMID 19660687
- [Background] Lopez-Soldado I, Avella M, Botham KM. Differential influence of different dietary fatty acids on very low-density lipoprotein secretion when delivered to hepatocytes in chylomicron remnants. Metabolism. 2009 Feb;58(2):186-95. doi: 10.1016/j.metabol.2008.09.012. PMID 19154951
- [Background] Deckelbaum RJ, Worgall TS, Seo T. n-3 fatty acids and gene expression. Am J Clin Nutr. 2006 Jun;83(6 Suppl):1520S-1525S. doi: 10.1093/ajcn/83.6.1520S. PMID 16841862
- [Background] Botham KM, Zheng X, Napolitano M, Avella M, Cavallari C, Rivabene R, Bravo E. The effects of dietary n-3 polyunsaturated fatty acids delivered in chylomicron remnants on the transcription of genes regulating synthesis and secretion of very-low-density lipoprotein by the liver: modulation by cellular oxidative state. Exp Biol Med (Maywood). 2003 Feb;228(2):143-51. doi: 10.1177/153537020322800203. PMID 12563020
- [Background] Mills SC, Windsor AC, Knight SC. The potential interactions between polyunsaturated fatty acids and colonic inflammatory processes. Clin Exp Immunol. 2005 Nov;142(2):216-28. doi: 10.1111/j.1365-2249.2005.02851.x. PMID 16232207
- [Background] Lalia AZ, Dasari S, Robinson MM, Abid H, Morse DM, Klaus KA, Lanza IR. Influence of omega-3 fatty acids on skeletal muscle protein metabolism and mitochondrial bioenergetics in older adults. Aging (Albany NY). 2017 Apr;9(4):1096-1129. doi: 10.18632/aging.101210. PMID 28379838
- [Background] Arterburn LM, Hall EB, Oken H. Distribution, interconversion, and dose response of n-3 fatty acids in humans. Am J Clin Nutr. 2006 Jun;83(6 Suppl):1467S-1476S. doi: 10.1093/ajcn/83.6.1467S. PMID 16841856
- [Background] von Schacky C, Weber PC. Metabolism and effects on platelet function of the purified eicosapentaenoic and docosahexaenoic acids in humans. J Clin Invest. 1985 Dec;76(6):2446-50. doi: 10.1172/JCI112261. PMID 3001149
- [Background] Khair-el-Din TA, Sicher SC, Vazquez MA, Wright WJ, Lu CY. Docosahexaenoic acid, a major constituent of fetal serum and fish oil diets, inhibits IFN gamma-induced Ia-expression by murine macrophages in vitro. J Immunol. 1995 Feb 1;154(3):1296-306. PMID 7822798
- [Background] Kostoglou-Athanassiou I, Athanassiou L, Athanassiou P. The Effect of Omega-3 Fatty Acids on Rheumatoid Arthritis. Mediterr J Rheumatol. 2020 Jun 30;31(2):190-194. doi: 10.31138/mjr.31.2.190. eCollection 2020 Jun. PMID 32676556
- [Background] Cicero AF, Ertek S, Borghi C. Omega-3 polyunsaturated fatty acids: their potential role in blood pressure prevention and management. Curr Vasc Pharmacol. 2009 Jul;7(3):330-7. doi: 10.2174/157016109788340659. PMID 19601857
- [Background] Ando, K., Watanabe, T., Daidoji, H., Otaki, Y., Hashimoto, N., Kumagai, Y., ... & Kubota, I. (2015). Combination therapy of eicosapentaenoic acid and pitavastatin for coronary plaque regression evaluated by integrated backscatter intravascular ultrasonography: a randomized controlled trial. Circulation, 132(suppl_3), A12007-A12007. https://doi.org/10.1161/circ.132.suppl_3.12007
- [Background] Mita T, Watada H, Ogihara T, Nomiyama T, Ogawa O, Kinoshita J, Shimizu T, Hirose T, Tanaka Y, Kawamori R. Eicosapentaenoic acid reduces the progression of carotid intima-media thickness in patients with type 2 diabetes. Atherosclerosis. 2007 Mar;191(1):162-7. doi: 10.1016/j.atherosclerosis.2006.03.005. Epub 2006 Apr 17. PMID 16616147
- [Background] Yoshiaki Shintani, Tomohiro Kawasaki, THE IMPACT OF A PURE-EPA OMEGA-3 FATTY ACID ON CORONARY PLAQUE STABILIZATION; A PLAQUE COMPONENT ANALYSIS WITH 64-SLICE MULTI-DETECTOR ROW COMPUTED TOMOGRAPHY, Journal of the American College of Cardiology, Volume 59, Issue 13, Supplement, 2012, Page E1731, ISSN 0735-1097, https://doi.org/10.1016/S0735-1097(12)61732-X. (https://www.sciencedirect.com/science/article/pii/S073510971261732X)
- [Background] Wakita, Yoshinori, Yasushi Wakida, Takahumi Itou, and Rika Mizuno. "High Purity Eicosapentaenoic Acid in Addition to a Strong Statin Makes Regression of Coronary Plaque in Patients with Angina Pectoris." (2011): A8893-A8893. https://www.ahajournals.org/doi/10.1161/circ.124.suppl_21.A8893
- [Background] Niki T, Wakatsuki T, Yamaguchi K, Taketani Y, Oeduka H, Kusunose K, Ise T, Iwase T, Yamada H, Soeki T, Sata M. Effects of the Addition of Eicosapentaenoic Acid to Strong Statin Therapy on Inflammatory Cytokines and Coronary Plaque Components Assessed by Integrated Backscatter Intravascular Ultrasound. Circ J. 2016;80(2):450-60. doi: 10.1253/circj.CJ-15-0813. Epub 2015 Dec 11. PMID 26667367
- [Background] Cawood AL, Ding R, Napper FL, Young RH, Williams JA, Ward MJ, Gudmundsen O, Vige R, Payne SP, Ye S, Shearman CP, Gallagher PJ, Grimble RF, Calder PC. Eicosapentaenoic acid (EPA) from highly concentrated n-3 fatty acid ethyl esters is incorporated into advanced atherosclerotic plaques and higher plaque EPA is associated with decreased plaque inflammation and increased stability. Atherosclerosis. 2010 Sep;212(1):252-9. doi: 10.1016/j.atherosclerosis.2010.05.022. Epub 2010 May 20. PMID 20542512
- [Background] Nishio R, Shinke T, Otake H, Nakagawa M, Nagoshi R, Inoue T, Kozuki A, Hariki H, Osue T, Taniguchi Y, Iwasaki M, Hiranuma N, Konishi A, Kinutani H, Shite J, Hirata K. Stabilizing effect of combined eicosapentaenoic acid and statin therapy on coronary thin-cap fibroatheroma. Atherosclerosis. 2014 May;234(1):114-9. doi: 10.1016/j.atherosclerosis.2014.02.025. Epub 2014 Mar 5. PMID 24637411
- [Background] Grenon SM, Aguado-Zuniga J, Hatton JP, Owens CD, Conte MS, Hughes-Fulford M. Effects of fatty acids on endothelial cells: inflammation and monocyte adhesion. J Surg Res. 2012 Sep;177(1):e35-43. doi: 10.1016/j.jss.2012.04.010. Epub 2012 Apr 27. PMID 22572621
- [Background] Combination Eicosapentaenoic Acid and Statin Treatment Reversed Endothelial Dysfunction in HUVECs Exposed to Oxidized LDL R. Preston Mason, PhD ∙ Robert F. Jacob, PhD ∙ J. Jose Corbalan, PhD ∙ Tadeusz Malinski, PhD
- [Background] Terano T, Shiina T, Tamura Y. Eicosapentaenoic acid suppressed the proliferation of vascular smooth muscle cells through modulation of various steps of growth signals. Lipids. 1996 Mar;31 Suppl:S301-4. doi: 10.1007/BF02637096. PMID 8729139
- [Background] McLennan PL. Myocardial membrane fatty acids and the antiarrhythmic actions of dietary fish oil in animal models. Lipids. 2001;36 Suppl:S111-4. doi: 10.1007/s11745-001-0692-x. PMID 11837983
- [Background] Mozaffarian D, Lemaitre RN, Kuller LH, Burke GL, Tracy RP, Siscovick DS; Cardiovascular Health Study. Cardiac benefits of fish consumption may depend on the type of fish meal consumed: the Cardiovascular Health Study. Circulation. 2003 Mar 18;107(10):1372-7. doi: 10.1161/01.cir.0000055315.79177.16. PMID 12642356
- [Background] Albert CM, Hennekens CH, O'Donnell CJ, Ajani UA, Carey VJ, Willett WC, Ruskin JN, Manson JE. Fish consumption and risk of sudden cardiac death. JAMA. 1998 Jan 7;279(1):23-8. doi: 10.1001/jama.279.1.23. PMID 9424039
- [Background] Siscovick DS, Raghunathan TE, King I, Weinmann S, Wicklund KG, Albright J, Bovbjerg V, Arbogast P, Smith H, Kushi LH, et al. Dietary intake and cell membrane levels of long-chain n-3 polyunsaturated fatty acids and the risk of primary cardiac arrest. JAMA. 1995 Nov 1;274(17):1363-7. doi: 10.1001/jama.1995.03530170043030. PMID 7563561
- [Background] Kang JX, Leaf A. Protective effects of free polyunsaturated fatty acids on arrhythmias induced by lysophosphatidylcholine or palmitoylcarnitine in neonatal rat cardiac myocytes. Eur J Pharmacol. 1996 Feb 15;297(1-2):97-106. doi: 10.1016/0014-2999(95)00701-6. PMID 8851173
- [Background] McLennan PL, Bridle TM, Abeywardena MY, Charnock JS. Dietary lipid modulation of ventricular fibrillation threshold in the marmoset monkey. Am Heart J. 1992 Jun;123(6):1555-61. doi: 10.1016/0002-8703(92)90809-a. PMID 1595535
- [Background] Kang JX, Xiao YF, Leaf A. Free, long-chain, polyunsaturated fatty acids reduce membrane electrical excitability in neonatal rat cardiac myocytes. Proc Natl Acad Sci U S A. 1995 Apr 25;92(9):3997-4001. doi: 10.1073/pnas.92.9.3997. PMID 7732020
- [Background] Murnaghan MF. Effect of fatty acids on the ventricular arrhythmia threshold in the isolated heart of the rabbit. Br J Pharmacol. 1981 Aug;73(4):909-15. doi: 10.1111/j.1476-5381.1981.tb08745.x. PMID 7272591
- [Background] Xiao YF, Gomez AM, Morgan JP, Lederer WJ, Leaf A. Suppression of voltage-gated L-type Ca2+ currents by polyunsaturated fatty acids in adult and neonatal rat ventricular myocytes. Proc Natl Acad Sci U S A. 1997 Apr 15;94(8):4182-7. doi: 10.1073/pnas.94.8.4182. PMID 9108126
- [Background] Xiao YF, Wright SN, Wang GK, Morgan JP, Leaf A. Fatty acids suppress voltage-gated Na+ currents in HEK293t cells transfected with the alpha-subunit of the human cardiac Na+ channel. Proc Natl Acad Sci U S A. 1998 Mar 3;95(5):2680-5. doi: 10.1073/pnas.95.5.2680. PMID 9482947
- [Background] Billman GE, Kang JX, Leaf A. Prevention of sudden cardiac death by dietary pure omega-3 polyunsaturated fatty acids in dogs. Circulation. 1999 May 11;99(18):2452-7. doi: 10.1161/01.cir.99.18.2452. PMID 10318669
- [Background] Kang JX, Leaf A. Antiarrhythmic effects of polyunsaturated fatty acids. Recent studies. Circulation. 1996 Oct 1;94(7):1774-80. doi: 10.1161/01.cir.94.7.1774. No abstract available. PMID 8840874
- [Background] Leaf, A. (2001). The electrophysiological basis for the antiarrhythmic actions of polyunsaturated fatty acids. European heart journal supplements, 3(suppl_D), D98-D105. https://doi.org/10.1016/S1520-765X(01)90127-0
- [Background] Jouven X, Charles MA, Desnos M, Ducimetiere P. Circulating nonesterified fatty acid level as a predictive risk factor for sudden death in the population. Circulation. 2001 Aug 14;104(7):756-61. doi: 10.1161/hc3201.094151. PMID 11502698
- [Background] Christensen JH. Omega-3 polyunsaturated Fatty acids and heart rate variability. Front Physiol. 2011 Nov 16;2:84. doi: 10.3389/fphys.2011.00084. eCollection 2011. PMID 22110443
- [Background] Thifault E, Cormier H, Bouchard-Mercier A, Rudkowska I, Paradis AM, Garneau V, Ouellette C, Lemieux S, Couture P, Vohl MC. Effects of age, sex, body mass index and APOE genotype on cardiovascular biomarker response to an n-3 polyunsaturated fatty acid supplementation. J Nutrigenet Nutrigenomics. 2013;6(2):73-82. doi: 10.1159/000350744. Epub 2013 May 8. PMID 23689286
- [Background] Harris WS. n-3 fatty acids and serum lipoproteins: human studies. Am J Clin Nutr. 1997 May;65(5 Suppl):1645S-1654S. doi: 10.1093/ajcn/65.5.1645S. PMID 9129504
- [Background] Nording ML, Yang J, Georgi K, Hegedus Karbowski C, German JB, Weiss RH, Hogg RJ, Trygg J, Hammock BD, Zivkovic AM. Individual variation in lipidomic profiles of healthy subjects in response to omega-3 Fatty acids. PLoS One. 2013 Oct 24;8(10):e76575. doi: 10.1371/journal.pone.0076575. eCollection 2013. PMID 24204640
- [Background] Mozaffarian D, Stein PK, Prineas RJ, Siscovick DS. Dietary fish and omega-3 fatty acid consumption and heart rate variability in US adults. Circulation. 2008 Mar 4;117(9):1130-7. doi: 10.1161/CIRCULATIONAHA.107.732826. Epub 2008 Feb 19. PMID 18285566
- [Background] Fabian CJ, Kimler BF, Hursting SD. Omega-3 fatty acids for breast cancer prevention and survivorship. Breast Cancer Res. 2015 May 4;17(1):62. doi: 10.1186/s13058-015-0571-6. PMID 25936773
- [Background] Bodkowski, R., Patkowska-Sokola, B., Filip-Psurska, B., Kempinska, K., Wietrzyk, J., Czyz, K., ... & Usydus, Z. (2014). Evaluation of the anti-proliferative activity of natural lipid preparations against tumor cell lines. J. Anim. Vet. Adv, 13(4), 257-266. DOI:10.3923/javaa.2014.257.266
- [Background] Tsao, C.S. An overview of ascorbic acid chemistry and biochemistry. In Vitamin C in Health and Disease; Packer, L., Fuchs, J., Eds.; Marcel Dekker Inc.: New York, NY, USA, 1997; pp. 25-58.
- [Background] Hamabe A, Takase B, Uehata A, Kurita A, Ohsuzu F, Tamai S. Impaired endothelium-dependent vasodilation in the brachial artery in variant angina pectoris and the effect of intravenous administration of vitamin C. Am J Cardiol. 2001 May 15;87(10):1154-9. doi: 10.1016/s0002-9149(01)01485-0. PMID 11356389
- [Background] Athanasiou A, Charalambous M, Anastasiou T, Aggeli K, Soteriades ES. Preoperative and postoperative administration of vitamin C in cardiac surgery patients - settings, dosages, duration, and clinical outcomes: a narrative review. Ann Med Surg (Lond). 2024 Apr 29;86(6):3591-3607. doi: 10.1097/MS9.0000000000002112. eCollection 2024 Jun. PMID 38846824
- [Background] Athanasiou A, Charalambous M, Anastasiou T, Soteriades ES. Pre- and post-operative administration of omega-3 polyunsaturated fatty acids in cardiac surgery patients. A narrative review. Ann Med Surg (Lond). 2025 Mar 18;87(4):2068-2092. doi: 10.1097/MS9.0000000000003061. eCollection 2025 Apr. PMID 40212170
- [Background] Ouagueni A, Shi Z, Shraim M, Al-Zoubi RM, Zarour A, Al-Ansari A, Bawadi H. Omega-3 Supplementation in Coronary Artery Bypass Graft Patients: Impact on ICU Stay and Hospital Stay-A Systematic Review and Meta-Analysis. Nutrients. 2024 Sep 29;16(19):3298. doi: 10.3390/nu16193298. PMID 39408265
- [Background] Howlett JG, Stebbins A, Petrie MC, Jhund PS, Castelvecchio S, Cherniavsky A, Sueta CA, Roy A, Pina IL, Wurm R, Drazner MH, Andersson B, Batlle C, Senni M, Chrzanowski L, Merkely B, Carson P, Desvigne-Nickens PM, Lee KL, Velazquez EJ, Al-Khalidi HR; STICH Trial Investigators. CABG Improves Outcomes in Patients With Ischemic Cardiomyopathy: 10-Year Follow-Up of the STICH Trial. JACC Heart Fail. 2019 Oct;7(10):878-887. doi: 10.1016/j.jchf.2019.04.018. Epub 2019 Sep 11. PMID 31521682
- See also: World Health Organization. (2014). Global status report on noncommunicable diseases 2014. WHO/NMH/NVI/15.1 World Health Organization. — https://www.who.int/publications/i/item/9789241564854
- See also: World Health Organization. (2021). Cardiovascular diseases (CVDs) factsheet. Updated June 2021. — https://www.who.int/news-room/fact-sheets/detail/cardiovascular-diseases-(cvds)
- See also: World Health Organization. (2003). Diet, nutrition and the prevention of chronic diseases : report of a joint WHO/FAO expert consultation, Geneva, 28 January - 1 February 2002. World Health Organization. — https://apps.who.int/iris/handle/10665/42665
- See also: Katoh, A., & Ikeda, H. (2011). Daily intake of eicosapentaenoic acid inhibits the progression of carotid intimal-media thickness in patients with dyslipidemia. Ther Res, 32(6), 863-8. — https://www.researchgate.net/publication/289048589_Daily_intake_of_eicosapentaenoic_acid_inhibits_the_progression_of_carotid_intimal-media_thickness_in_patients_with_dyslipidemia
- See also: Doherty, W. O. S., Mousavioun, P., & Fellows, C. M. (2011). Value-adding to cellulosic ethanol: Lignin polymers. Industrial Crops and Products, 33(2), 259-276. — https://doi.org/10.1016/j.indcrop.2010.10.022